


## **Statistical Analysis Plan**

#### Version 1

TITLE: 99mTc-rhAnnexin V-128 Imaging of Apoptosis and Cardiotoxicity in Relationship to Ventricular Function in Patients with Early Stage Breast Cancer Receiving Doxorubicin-Based Chemotherapy

PROTOCOL #: AAA-Annexin-05 v.7.0 dated 11 March 2018

NCT #: NCT02677714

PHASE: Proof of Concept and Phase II study

DATE: Final version 1 dated 22 March 2019

DESIGN: Single centre study.

INVESTIGATIONAL PRODUCT: Kit for the Preparation of Tc-99m Recombinant Human Annexin V-128 for Injection




Version: 021 Page: **2 of 96** 

### **APPROVAL/REVISION HISTORY**

#### Autorship/Approval



#### **Revision history**

| Rev. | Name | Date | Note |
|------|------|------|------|
| 1 | | | |

#### Sent to

| Rev. | Name | e-mail | Sent on | Note |
|------|------|--------|---------|------|
| 01 | | | | |


Version: 021 Page: **3 of 96** 

## 1 Index

| 1 | Index | 3 |
|---|---|---|
| 2 | List of abbreviations | 8 |
| 3 | Protocol title and number | 11 |
| 4 | INFORMATION TAKEN FROM THE PROTOCOL | 12 |
| | 4.1 Study objectives | 12 |
| | 4.1.1 Primary objective | |
| | 4.1.2 Secondary objective | |
| | 4.2 Study design | 13 |
| | 4.2.1 Study population | |
| | 4.2.1.2 Exclusion criteria | 14 |
| | 4.2.2 Study exposure | |
| | 4.3 Methods and procedures | |
| | 4.3.1 Source of study population | 15<br>15 |
| | 4.3.3.2 Efficacy assessments | 16 |
| | 4.3.3.2.1 <sup>99m</sup> Tc-rhAnnexin V-128 SPECT imaging and image analysis | 16 |
| | 4.3.3.2.2 Cardiac magnetic resonance imaging | 16 |
| | 4.3.3.2.3 Cardiotoxicity biomarkers assessments | 17 |
| | 4.3.3.3 Safety assessments | 17 |
| | 4.3.3.3.1 Adverse events and other safety aspects | 18 |
| | 4.3.3.3.2 Laboratory assessments | 19 |
| | 4.3.3.3.3 Immunogenicity assessments | 20 |
| | 4.3.3.3.4 Radiation risk assessment | 20 |
| | 4.3.3.4 Withdrawal/discontinuation | 20 |
| | 4.3.3.5 Prohibitions and restrictions | 21 |


| | | | Version: 021 Page | e: <b>4 of 9</b> 6 |
|---|---|---|---|---|
| | 4.3.4 | Schedule | of assessments | 21 |
| | 4.3.5 | Planned | sample size | 23 |
| 5 | SUBJEC | T POPUL | ATIONS (ANALYSIS SETS) | 25 |
| | 5.1 Effic | сасу | | 25 |
| | 5.1.1 | Full analy | /sis set (FAS) | 25 |
| | 5.1.2 | Per Proto | ocol population (PP) | 25 |
| | 5.2 Safe | ety set | | 25 |
| | 5.3 Prin | nary popul | ation | 25 |
| 6 | STATIST | TICAL ME | THODS | 26 |
| | 6.1 Stat | tistical ana | lysis strategy | 26 |
| | 6.1.1 | Efficacy | endpoint(s) | 26 |
| | 6.1. | | ary endpoint of PoC | |
| | 6.1. | .1.2 Prim | ary endpoint of Phase II | 26 |
| | 6.1. | .1.3 Seco | ondary endpoints | 26 |
| | | = | ndpoint(s) | |
| | | | erse events | |
| | 6.1. | | cal laboratory values | |
| | 6.1. | | signs and medical review | |
| | 6.1.3<br>6.1. | • | lata and outliersing data | |
| | | | ing or incomplete dates | |
| | 6.1.<br>6.1. | | ers | |
| | | | lisposition | |
| | 6.1.4<br>6.1.5 | • | rals | |
| | 6.1.6 | | phic and baseline characteristics | |
| | 6.1.7 | | and surgical history | |
| | 6.1.8 | | compliance | |
| | 6.1.9<br>6.1.10 | | concomitant therapieslata | |
| | | | lows | |
| | | | d data formats | |
| | | | of centres | |
| | | | nalysis | |
| | | | dependent data monitoring committee (DMC) / interim data review committee | |
| | | | es and analysis of subgroupsy analysisy | |
| | | | y | |
| | | | nce testing and estimation | |
| 7 | COMPU | TER SYST | EMS, SOFTWARE AND VALIDATION OF PROGRAMS | 33 |


| | | Version: 021 | Page: <b>5 of 96</b> |
|---|---|---|---|
| 7.1 | Hardware | | 33 |
| 7.2 | Software | | 33 |
| 7.3 | Validation | programs | 33 |
| 8 CH | ANGES FR | OM PROTOCOL | 34 |
| 9 REI | FERENCES | 3 | 35 |
| 10 DA | TA PRESEN | NTATION | 36 |
| 10.1 | Listings in | dex | 36 |
| 10.2 | Listing tem | nplates | 37 |
| 10.3 | Tables ind | ex | 37 |
| 10.4 | Table tem | plates | 39 |
| 10.5 | Figures inc | dex | 39 |
| 10.6 | Figure tem | nplates | 40 |
| 10.7 | Statistical | appendix | 40 |
| 11 APF | PENDICES. | | 42 |
| 11.1 | Standard I | istings | 42 |
| Listing | 16.2.1.1: | Subject Disposition – All subjects | 43 |
| Listing | 16.2.1.2: | Subject Disposition – Study Withdrawals | 44 |
| Listing | 16.2.1.3: | Inclusion Criteria | 45 |
| Listing | 16.2.1.4: | Exclusion Criteria | 46 |
| Listing | 16.2.1.5: | Screening Failures | 47 |
| Listing | 16.2.2: | Protocol Deviations and Reasons for Exclusion from the Study Populations | 48 |
| Listing | 16.2.4.1: | Demographics | 49 |
| Listing | 16.2.4.2: | Medical History and Associated Pathologies | 50 |
| Listing | 16.2.4.3/1: | Prior and Concomitant Medications | 51 |
| Listing | 16.2.4.3/2: | Prior and Concomitant Medications | 52 |
| Listing | 16.2.5.1/1: | Study Drug Administration and Extent of Subject Exposure | 53 |


| | Version: 021 | Page: <b>6 of 96</b> |
|---|---|---|
| Listing 16.2.5.1/2: | Study Drug Administration and Extent of Subject Exposure | 54 |
| Listing 16.2.5.2: | Chemotherapy Treatment | 55 |
| Listing 16.2.6.1/1: | Imaging Assessment | 56 |
| Listing 16.2.6.1/2: | Imaging Assessment | 57 |
| Listing 16.2.6.2: | Cardiac Magnetic Resonance Imaging | 58 |
| Listing 16.2.6.3: | Cardiotoxicity Biomarkers | 59 |
| Listing 16.2.7.1/1: | All Adverse Events | 60 |
| Listing 16.2.7.1/2: | All Adverse Events | 61 |
| Listing 16.2.7.1/3: | All Adverse Events | 62 |
| Listing 16.2.7.2/1: | Serious Adverse Events | 63 |
| Listing 16.2.7.2/2: | Serious Adverse Events | 64 |
| Listing 16.2.7.2/3: | Serious Adverse Events | 65 |
| Listing 16.2.7.3/1: | Adverse Events Leading to Withdrawal | 66 |
| Listing 16.2.7.3/2: | Adverse Events Leading to Withdrawal | 67 |
| Listing 16.2.7.3/3: | Adverse Events Leading to Withdrawal | 68 |
| Listing 16.2.7.4/1: | Adverse Events with Outcome Death | 69 |
| Listing 16.2.7.4/2: | Adverse Events with Outcome Death | 70 |
| Listing 16.2.7.4/3: | Adverse Events with Outcome Death | 71 |
| Listing 16.2.8.1/1: | Hematology | 72 |
| Listing 16.2.8.2/1: | Blood Chemistry | 73 |
| Listing 16.2.8.3/1: | Urinalysis | 74 |
| Listing 16.2.8.4: | Immunogenicity | 75 |
| Listing 16.2.9.1: | Pregnancy Test | 76 |
| Listing 16.2.9.3: | Physical Examination | 77 |
| Listing 16.2.9.4: | Vital Signs | 78 |
| 11.2 Standard | Tables | 79 |



| | Version: 021 | Page: <b>7 of 9</b> 6 |
|---|---|---|
| Table 14.1.1: Subje | ect disposition | 80 |
| Table 14.1.4.1: De | mographics – FAS Population | 81 |
| Table 14.1.7.2/1: | Study Drug Administration – Safety Population | 82 |
| Table 14.1.7.2/2: | Study Drug Administration – Safety Population | 83 |
| Table 14.1.7.2/3: | Study Drug Administration – Safety Population | 84 |
| Table 14.3.1.1: Ov | rerall Summary of Adverse Events – Safety Population | 85 |
| | mber (%) of Subjects Reporting Treatment Emergent Adverse Events<br>and Preferred Term – Safety Population | |
| Table 14.3.1.3: Nu<br>Safety Population 87 | mber (%) of Subjects Reporting Treatment Emergent Adverse Events b | y Severity – |
| | mber (%) of Subjects Reporting Treatment Emergent Adverse Drug Fulation | |
| | mber (%) of Subjects Reporting Treatment Emergent Serious Advers<br>n Class and Preferred Term – Safety Population | |
| | mber (%) of Subjects Reporting Treatment Emergent Serious Advers | |
| | mber (%) of Subjects Reporting Treatment Emergent Serious Adverse Dropulation | |
| Table 14.3.2.1: Lis | ting of Adverse Events with Outcome Death – Safety Population | 92 |
| Table 14.3.2.2: Lis | ting of Serious Adverse Events – Safety Population | 93 |
| 11.3 Standard Figu | ıres | 94 |
| 12 APPENDICES TO | THE SAP TEMPLATE | 95 |
| 12.1 Derived data | | 95 |
| 12.2 SAS programs | S | 96 |



Version: 021 

#### 2 List of abbreviations

AAA Advanced Accelerator Applications

AC Doxorubicin/Cyclophosphamide chemotherapy

AE Adverse Event

ALAT Alanine Aminotransferase

ALP Alkanine Phosphatase

ALT Alanine Transaminase

ANOVA ANalysis Of VAriance

ASAT Aspartate Aminotransferase

AST Aspartate Transaminase

ATC Anatomical Therapeutic Chemical classification system

AU Absolute Uptake

BMI Body Mass Index

BP Blood Pressure

C.I. Confidence Interval

CMRI Cardiac Magnetic Resonance Imaging

CRF Case Report Form

CRO Clinical Research Organization

CT Computed Tomography

CTCAE Common Terminology Criteria for Adverse Events

CUR Cardiac Uptake Ratio

DMC Data Monitoring Committee

DSMB Data Safety Monitoring Board

ECOG Eastern Cooperative Oncology Group

eCRF Electronic Case Report Form

ELISA Enzyme-Linked ImmunoSorbent Assay

FAS Full Analysis Set

GCP Good Clinical Practice

GGT Gamma-Glutamyl Transpeptidase


Version: 021 Page: **9 of 96** 

Hb Hemoglobin

HR Heart Rate

ICF Informed Consent Form

ICH International Conference on Harmonization

ID Identification

ID/gInjected Dose per gramIPInvestigational Product

IQR Interquartile Range

ITT Intention To Treat

kVp Peak Kilovoltage

LGE Late gadolinium enhancement

LLT Lowest Level Term

LV Left Ventricular

LVEF Left Ventricular Ejection Fraction

MBq Mega Becquerel

MCV Mean Corpuscular Volume

MHLTC Ministry of Health and Long Term Care

MedDRA Medical Dictionary for Regulatory Activities

MRI Magnetic Resonance Imaging

NCI National Cancer Institute

NT-proBNP N Terminal pro B-type Natriuretic Peptide

OHSN-REB Ottawa Hospital Science Network Research Ethics Board

PoC Proof of Concept

PP Per Protocol

PT Preferred Term

RBC Red Blood Cells

REB Research Ethic Board

ROI Region of Interest

SAE Serious Adverse Event


Version: 021  SAP Statistical Analysis Plan S.D. Standard Deviation SOC System Organ Class Single-Photon Emission Computed Tomography SPECT Standardized Uptake Value SUV Echo Time ΤE TR Repetition Time University of Ottawa Heart Institute UOHI

White Blood Cells

**WBC** 


Version: 021 Page: **11 of 96** 

#### 3 Protocol title and number

<sup>99m</sup>Tc-rhAnnexin V-128 Imaging of Apoptosis and Cardiotoxicity in Relationship to Ventricular Function in Patients with Early Stage Breast Cancer Receiving Doxorubicin-Based Chemotherapy (Protocol Number AAA-Annexin-05 v.7.0 dated 11 March 2018).




Version: 021 Page: **12 of 96** 

#### 4 INFORMATION TAKEN FROM THE PROTOCOL

#### 4.1 Study objectives

#### 4.1.1 Primary objective

The primary objective of this study is to investigate <sup>99m</sup>Tc-rhAnnexin V-128 imaging of apoptosis in the evaluation of doxorubicin-induced cardiotoxicity in patients with early stage breast cancer.

#### 4.1.1.1 Primary hypothesis

Patients with early stage breast cancer undergoing doxorubicin-containing (neo) adjuvant chemotherapy will have increased uptake of <sup>99m</sup>Tc-rhAnnexin V-128 at the end of the 2<sup>nd</sup> and the 4<sup>th</sup> cycles of AC treatment, and 12 weeks after the last cycle of doxorubicin, compared to baseline uptake.

#### 4.1.2 Secondary objective

The secondary objectives of this study are:

- To determine the timing and extent of <sup>99m</sup>Tc-rhAnnexin V-128 imaging of apoptosis (<sup>99m</sup>Tc-rhAnnexin V-128 myocardial uptake).
- To determine the relationship between <sup>99m</sup>Tc-rhAnnexin V-128 myocardial uptake and the changes in left ventricular (LV) function measured by cardiac magnetic resonance imaging (CMRI) and the changes in the cardiotoxicity biomarkers.

#### 4.1.2.1 Secondary hypotheses

- Patients with early stage breast cancer undergoing doxorubicin-containing (neo) adjuvant chemotherapy will have worsening of LV function measured with CMRI at the end of the 2<sup>nd</sup> and the 4<sup>th</sup> cycle of treatment and 12 weeks from the last dose of doxorubicin chemotherapy compared to baseline.
- The uptake of <sup>99m</sup>Tc-rhAnnexin V-128 (percentage of injected dose per gram, % ID/g) will correlate with changes in CMRI LV function parameters and changes in the cardiotoxicity biomarkers.




on: 021 Page: **13 of 96** 

#### 4.2 Study design

This is a single centre, Proof of Concept (PoC), Phase II study. Patients with histologically confirmed early stage (Stage I, II and III) HER-2 negative breast cancer and scheduled to receive (neo) adjuvant doxorubicin-based chemotherapy (A - 60 mg/m²; C - 600 mg/m²; every 2 or 3 weeks x 4 cycles) to be followed by paclitaxel or docetaxel as per clinical practice will be recruited from the Ottawa Hospital Cancer Centre. Participants will be scheduled for cardiac MRI and <sup>99m</sup>Tc-rhAnnexin V-128 imaging prior to initiating doxorubicin-based chemotherapy. Participants will also undergo <sup>99m</sup>Tc-rhAnnexin V-128 imaging and CMRI at the end of the 2<sup>nd</sup> and the 4<sup>th</sup> cycles of AC treatment and 12 weeks after the last cycle.

#### 4.2.1 Study population

Approval for the study will be obtained from the Ottawa Hospital Science Network Research Ethics Board (OHSN-REB) and Health Canada. All participants will provide written informed consent prior to the initiation of any study procedures. It is foreseen to recruit thirty patients with early stage breast cancer.

#### 4.2.1.1 Inclusion criteria

- Females ≥ 18 years of age with histologically confirmed early stage (stage I, II or III) HER-2 negative breast cancer and planned to receive (neo) adjuvant doxorubicin-based (A 60 mg/m²; C 600 mg/m²; every 2 or 3 weeks x 4 cycles) chemotherapy.
- 2. Eastern Cooperative Oncology Group Status (ECOG) ≤ 2 (see Appendix II of study protocol).
- 3. Able and willing to comply with the study procedures.




Version: 021 Page: **14 of 96** 

#### 4.2.1.2 Exclusion criteria

- 1. Pregnancy or lactation.
- 2. Moderate or severe valvular stenosis or regurgitation.
- 3. History of atrial fibrillation or flutter.
- 4. History of any disease or relevant physical or psychiatric condition which may interfere with the study objectives at the investigator judgment.
- 5. Known hypersensitivity to the investigational product or any of its components.
- 6. Prosthetic valve or pacemaker.
- 7. Claustrophobia or inability to lie still in a supine position.
- 8. Contraindication(s) to CMRI procedure.
- 9. Participation in another clinical trial within 4 weeks before study inclusion, except for patients who have participated or who are currently participating in a study without any study drug administration.
- 10. Unwillingness to provide consent.

#### 4.2.2 Study exposure

The "Kit for preparation of <sup>99m</sup>Tc-rhAnnexin V-128 for injection" consists of 1 dose. Participants will receive 1 dose of 350 MBq ± 10% of <sup>99m</sup>Tc-rhAnnexin V-128 administered as a single intravenous bolus over 10-20 seconds at each of the four MRI scans (at screening, after the 2<sup>nd</sup> cycle, after the 4<sup>th</sup> cycle and 12 weeks after AC chemotherapy). Thus subjects will be exposed to a total of 4 <sup>99m</sup>Tc-rhAnnexin V-128 injections.

#### 4.2.3 Termination of the study

Early termination of the study can occur in the following cases:

- When the visual review and analysis of the images of the first 10 participants by the DMC does not demonstrate the diagnostic potential of the study product in terms of quality or efficacy, the Sponsor may discontinue the clinical study by sending a written notice to the investigator and competent authorities.
- When the Sponsor is aware of new information on matters concerning the safety of the study
  product, as well as other important information that may affect proper conduct of the clinical
  study, the Sponsor may discontinue the clinical study and send a written notice of the
  discontinuation to the investigator and competent authorities.
- If the investigator intends to discontinue participation in the study, the investigator must immediately inform the Sponsor in written about the discontinuation and the reason for it.




Version: 021 Page: **15 of 96** 

The study is stopped by a regulatory authority.

If none of the previous condition applies, the end of study is defined as the completion of all study procedures in the last enrolled participant (i.e. last visit, last participant).

The Sponsor reserves the right to discontinue the study at any time for any reason by sending a written notice of the discontinuation to the investigator and competent authorities.

#### 4.3 Methods and procedures

#### 4.3.1 Source of study population

Patients from the Ottawa Hospital Cancer Centre will be enrolled. The Ottawa Hospital Cancer Centre sees about 1,000 patients per year with breast cancer (Stage I to III) and it is estimated that 4 to 5 per month would meet the study inclusion criteria. We plan to recruit 30 patients over 18 to 24 months, or approximately 1 to 2 patients per month.

#### 4.3.2 Participant study identification

A unique participant identification number (Participant ID) will be assigned at the start of the screening period to each participant who signs the informed consent form. This number will identify the participant throughout the study. Participant IDs will include the 2-digit protocol number (05), the 2-letter code (CA) and a 3-digit participant number (ex: 05-CA-001 for first participant in).

#### 4.3.3 Study procedure

Voluntary written informed consent will be obtained prior to the initiation of any study-related procedures. Study conduct procedures will include a screening visit and the imaging visits.

#### 4.3.3.1 Baseline assessments

- Each participant's date of birth (mm/yyyy), gender, ethnicity, medical history, and relevant baseline characteristics will be recorded.
- Inclusion and Exclusion criteria will be checked.
- Results from any standard of care testing related to the participant's condition will be collected and will include baseline echocardiography when available.
- Women of childbearing potential must have negative pregnancy test at screening.
- Height, weight, BMI and vital signs will be recorded.




Version: 021 Page: **16 of 96** 

#### 4.3.3.2 Efficacy assessments

#### 4.3.3.2.1 99mTc-rhAnnexin V-128 Planar and SPECT imaging and image analysis

Administration of the <sup>99m</sup>Tc-rhAnnexin V-128 (350 MBq ± 10%) will be as a single bolus via an intravenous catheter in an antecubital vein followed by a saline flush. All images will be acquired with a dual head SPECT/CT gamma camera with low-energy high-resolution collimators. The energy acceptance window for the <sup>99m</sup>Tc photopeak will be 140 keV (± 10%). A low dose CT scan (helical, 120 kVp, 1 mA with 1.9 pitch) will be acquired of the thorax for attenuation correction.

Planar imaging will be performed in the anterior view with acquisition using a 256 x 256 matrix, an energy window set for Tc<sup>99m</sup> at 140 keV +/- 10% and a low energy, high resolution (LEHR) collimator. The image will be acquired for 1200s at one and two hours post injection of radiotracer.

Reconstruction will be done using iterative reconstruction incorporating CT-based attenuation correction and dual-energy-window scatter correction. Planar and SPECT images of the thorax will be acquired at 1 and 2 hours post injection. Acquired images will be stored for off-line analysis using a Hermes Gold workstation (Hermes Medical Solutions). Myocardial uptake will be measured from regions of interest (ROIs) placed over the myocardium on the SPECT images co-registered with the corresponding CT images for anatomic delineation. Myocardial uptake will be expressed in absolute units (% injected dose/g) or as a standardized uptake value (SUV). As a secondary analysis, a simpler approach without attenuation and scatter corrections will also be used by determination of a cardiac uptake ratio (CUR) with a second group of ROIs placed over the axillary soft tissues to obtain a value representative of background.

Inter and intra-observer variability will be determined by repeated analysis of the images of all participants.

#### 4.3.3.2.2 Cardiac magnetic resonance imaging

Cardiac MRI will be performed either with a 1.5-T scanner (Siemens, Erlangen, Germany) or a 3.0-T Scanner (Siemens, Erlangen, Germany). Transverse images will be acquired with an inversion recovery prepared dark blood HASTE sequence (repetition time [TR] 600 ms, echo time [TE] 26 ms, 6 mm slice thickness, 1.8 mm interslice gap, matrix 256x104). Cine bright-blood images in the 4-and 2-chamber and long-axis planes will be performed with a breath-hold balanced steady-state free precession sequence (true fast imaging with steady-state precession, TR 42 ms, TE 1.2 ms, flip





angle 70°, 6 mm slice thickness, matrix 192x174). Cine breath-hold balanced steady-state free precession short-axis images will be acquired for the entire LV from the base to the apex (stack of 10 sequential short-axis slices; TR 64 ms, TE 1 ms, flip angle 80°, 8 mm slice thickness, 1.6 mm interslice gap, matrix 192x132) to obtain measurements of left ventricular ejection fraction.

To evaluate for myocardial edema, dark blood T2-weighted turbo spin echo short-axis images will be obtained (TR 1,800 to 2,100 ms, TE 74 ms, 8 mm slice thickness, 4 mm interslice gap, matrix 256x175). At each imaging session, a single 5 mL blood sample will be withdrawn for measurement of the hematocrit, to be used in conjunction with the T1 measurements to ensure accurate estimation of extracellular volume. T1 maps in short-axis oblique and four chamber views using a modified Look-Locker inversion recovery, "MOLLI" will be acquired before the administration of contrast to obtain native T1 values. Late gadolinium enhancement (LGE) images will be obtained after 10 min of 0.2 mmol/kg injection of gadolinium (Gadovist®, Bayer Inc.) with a T1-weighted inversion recoveryprepared multislice true fast imaging with steady-state precession sequence with magnitude and phase-sensitive reconstruction. Images will be acquired sequentially in the short axis, followed by horizontal and vertical long-axis images (TR 700 ms, TE 1.0 ms, flip angle 40°, 8 mm slice thickness, 1.6 mm interslice gap, matrix 192x144). To quantify the myocardial mass of the LGE, the endocardial and epicardial borders of the short-axis view of the LV will be manually traced. The computerassisted detection algorithm will be used to define LGE as any region with a signal intensity ± 2 SD above a reference remote myocardial region. The LGE mass will be expressed as a percentage of the LV mass. 15 minutes post injection, we will acquire post contrast T1 maps in short-axis oblique and four chamber views. All analysis including quantitative will be performed with dedicated computer software (CVI 42, Circle Cardiovascular Imaging, Calgary, Alberta, Canada).

#### 4.3.3.2.3 Cardiotoxicity biomarkers assessments

Blood samples (3 mL) for cardiotoxicity biomarkers assessments (troponin, NT-proBNP) will also be collected at screening and before each injection of <sup>99m</sup>Tc-rhAnnexin V-128.

#### 4.3.3.3 Safety assessments

- Medical review, including the measurement of the weight and BMI, will be performed before each <sup>99m</sup>Tc-rhAnnexin V-128 administration.
- Measurement of vital signs (systolic and diastolic blood pressure and heart rate) will be performed 15 minutes before each <sup>99m</sup>Tc-rhAnnexin V-128 administration and at the end of the second imaging procedure.



Version: 021 Page: **18 of 96** 

- Women of childbearing potential must have negative pregnancy test at screening, before each IP administration and before each CMRI (in case the CMRI is not performed on the same day of IP administration).
- After signature of the ICF, any medical events defined as Adverse Events will be recorded and followed until the last study related procedure or until resolution.
- All medications taken from 2 weeks prior to the first administration date through the end of study will be recorded as concomitant medications.

#### 4.3.3.3.1 Adverse events and other safety aspects

#### **Definition of Adverse Events**

An AE is defined as any untoward medical occurrence in a participant and which does not necessarily have a causal relationship with the IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal clinically significant laboratory finding), symptom, or disease, temporarily associated with the use of an IP, whether or not causally related to the IP.

AEs will be reported, if applicable, from the signing of the informed consent until the last study-related procedure. AE severity will be assessed according to the grading system of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE) as included in Appendix III of study protocol.

#### **Definition of Serious Adverse Events**

A SAE is any untoward medical occurrence that at any dose:

- results in death;
- is life-threatening;
  - Note: "life-threatening" refers to an event in which the participant is at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it was more severe;
- results in persistent or significant disability/incapacity;
- results in congenital anomaly or birth defect;
- requires in-participant hospitalization or leads to prolongation of hospitalization, with the exception of elective pre-planned hospitalizations.

Serious Adverse Events (SAE) will be defined according to ICH/GCP and Regulatory Standards. SAEs will be reported from the signing of the informed consent and followed until resolution or determined to be not clinically significant. The specific SAE Reporting Form should be used (Appendix IV of study protocol).




Version: 021 Page: **19 of 96** 

#### Procedure in Case of Pregnancy

Prior to clinical study enrolment, women of childbearing potential must be advised of the importance of avoiding pregnancy during clinical study participation and the potential risks for an unintentional pregnancy. During the clinical study, all women of childbearing potential should use of a reliable means of contraception, and should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g. missed or late menstrual period).

The investigator must report to the Sponsor any pregnancy associated with IP exposure including conceptions occurring until 30 days after the IP administration using the specific Pregnancy Form (Appendix V of study protocol). Appropriate pregnancy follow-up procedures will be considered if indicated. The Investigator should respond in accordance with the reporting procedure for SAEs including information regarding the outcome of pregnancy.

#### New Safety Information Affecting the Conduct of the Study

Any information or changes significantly affecting the conduct of the trial and/or increasing the risk to participants will be provided to all investigators, REB(s), and Regulatory Authorities. Depending on the nature of the information or the changes, the protocol and/or the participant information may necessitate an amendment.

#### Data Monitoring and Safety

The data collected for this study is observational in design and will not be used for clinical care or clinical decision making. No formal DSMB will be formed. However, the safety data will be part of the review and assessment by the DMC.

#### 4.3.3.3.2 Laboratory assessments

Blood samples for hematology, blood chemistry and urinalysis will be obtained at baseline for screening, and 12 weeks after the end of chemotherapy and following any adverse effects attributed to the study procedures. Results from laboratory analysis conducted during the oncology treatment will be used for research analysis.

In the case of clinically significant abnormalities in baseline laboratory values, the participant will be declared as a screening failure.

| Hematology | Blood chemistry | Urinalysis |
|---|---|---|
| <ul> <li>WBC with differential</li> <li>RBC</li> <li>Platelets</li> <li>Hb</li> <li>MCV</li> <li>Hematocrit<sup>2</sup></li> </ul> | <ul> <li>Total bilirubin</li> <li>ALP</li> <li>AST/ASAT</li> <li>ALT/ALAT</li> <li>Gamma-GT</li> <li>Creatinine<sup>3</sup></li> </ul> | <ul> <li>Dipstick test<sup>1</sup></li> <li>Pregnancy test (at screening, before each injection of study product</li> </ul> |

# Statistical Analysis Plan ANNEXIN 05 Confidential Version: 021  and before each CMRI, if applicable)

Laboratory Assessments, including cardiotoxicity biomarkers assessments, will be performed at The Ottawa Hospital according to Ministry of Health and Long Term Care (MHLTC) standards.

#### 4.3.3.3 Immunogenicity assessments

Anti-rhAnnexin V-128 IgG and IgM antibodies will be quantified in serum samples by ELISA. For this purpose 10 mL blood samples will be collected at screening and 12 weeks after the last dose of doxorubicin, before injection of <sup>99m</sup>Tc-rhAnnexin V-128. Serum will be prepared, divided into six aliquots and frozen (-80°C). Three out of six serum samples per time-point will be shipped to the central laboratory \_\_\_\_\_\_\_. Remaining samples will be shipped only if required for analysis and destroyed at study end if not required.

#### 4.3.3.3.4 Radiation risk assessment

Participants will receive radiation from  $^{99m}$ Tc-rhAnnexin V-128 (350 MBq) for a dose of 3.0 mSv (8.1  $\pm$  0.8  $\mu$ Sv/MBq and from the CT scan for attenuation correction for a dose of 0.4 mSv. Total dose for the  $^{99m}$ Tc-rhAnnexin V-128 and CT will be 3.4 mSv for one imaging study and 13.6 mSv for the 4 administrations.

Since the annual background radiation dose at sea level in North America is 2.7 mSv, the total effect of dose for this study per patient radiation is equivalent to living 5 years in North America. This poses minimal risk to the participant and there are no expected consequences with this exposure.

#### 4.3.3.4 Withdrawal/discontinuation

The withdrawal of a study participant is mandatory in the following cases:

- Pregnancy
- Protocol violation determined as critical

<sup>&</sup>lt;sup>1</sup> If any of the assessments of the dipstick test is positive, a microscopic analysis of the urine must be performed.

<sup>&</sup>lt;sup>2</sup> An additional 5 mL blood sample will be collected at each CMRI visit for measurement of hematocrit to be used in conjunction with the T1 measurements to ensure accurate estimation of extracellular volume.

<sup>&</sup>lt;sup>3</sup> Creatinine will be repeated for CMRI when required if not clinically available.



Version: 021 Page: **21 of 96** 

- Lost to follow-up
- Serious intercurrent illness or other safety reasons for which the Investigator considers it is
  in the best interest of the participant to withdraw from the study
- Screening failure
- Failure to complete prescribed cycle of anthracycline chemotherapy

A "screening failure" is a participant who has signed the informed consent, but who does not meet all selection criteria following the screening evaluations. For participants not considered eligible after the screening period, the reason for not being eligible must be documented. No additional assessments are needed. Participant information collected at the Screening visit will be entered in the eCRF and will be used in the study analysis.

A participant may withdraw from the study at any time. The primary reason for a participant's withdrawal from the study should be determined if possible. The date and reason for discontinuation will be documented in the eCRF.

#### 4.3.3.5 Prohibitions and restrictions

Patients who are pregnant will not be permitted to participate in the study. Pregnancy tests will be performed for all study participants (of childbearing potential) at baseline and prior to each IP administration.

All imaging will be performed in an ambulatory care setting. There are no specific precautions required for participants upon completion of Annexin and CMR imaging.

Any concomitant medication deemed necessary for the welfare of the participant during the study may be given at the discretion of the Investigator. However, it is the responsibility of the Investigator to ensure that details regarding the medication are recorded in full in the case report form, including any changes that have occurred during the study.

#### 4.3.4 Schedule of assessments

Patients who have signed the informed consent and are eligible to participate in the study will undergo the following assessments:

• Screening will be conducted within 2 weeks prior to chemotherapy treatment initiation. Eligible and consenting patients will undergo a medical review (including measurement of the height, weight, and BMI), vital signs (systolic and diastolic blood pressure, heart rate), blood analysis and urinalysis. The following blood analysis will be conducted: cardiotoxicity biomarkers troponin and NT-proBNP (N terminal pro B-type natriuretic peptide), assessment



Version: 021 Page: **22 of 96** 

of anti-annexin V-128 antibodies (baseline value) and hematology/biochemistry as detailed in Section 4.3.3.3.2. Participants will undergo the first CMRI and SPECT/CT <sup>99m</sup>Tc-rhAnnexin V-128 scans.

- The planned chemotherapy treatment consists of doxorubicin 60 mg/m2 in combination with cyclophosphamide 600 mg/m2 IV (AC) every 2 or 3 weeks for 4 cycles to be followed by paclitaxel or docetaxel as per clinical practice, at the Ottawa General Hospital, with potential dose adjustments.
- After the 2<sup>nd</sup> cycle of doxorubicin and before the 3<sup>rd</sup> cycle, the participants will undergo a second series of study imaging procedures (CMRI, planar and SPECT/CT with <sup>99m</sup>Tc-rhAnnexin V-128). Blood sampling will be performed for the assessment of cardiotoxicity biomarkers (troponin, NT-proBNP).
- After the 4<sup>th</sup> cycle of doxorubicin and with 2 weeks after the 4<sup>th</sup> cycle, participants will undergo the third series of study imaging procedures (CMRI, planar and SPECT/CT with <sup>99m</sup>Tc-rhAnnexin V-128). Blood sampling will be performed for the assessment of cardiotoxicity biomarkers (troponin, NT-proBNP).
- At 12 weeks after the 4<sup>th</sup> cycle of doxorubicin, participants will undergo the fourth series of study imaging procedures (CMRI, planar and SPECT/CT with <sup>99m</sup>Tc-rhAnnexin V-128). Blood sampling will be performed for the assessment of cardiotoxicity biomarkers (troponin, NT-proBNP) and hematology/biochemistry as detailed in Section 4.3.3.3.2. Urinalysis will also be performed. Immunology blood sampling will be performed to rule out the development of anti-annexin V-128 antibodies.
- The imaging procedures will be conducted at the University of Ottawa Heart Institute (UOHI).
   Safety assessments will be done at each procedure. The CMRI and the SPECT/CT imaging will be done on the same day or within one week of each other.
- Relevant results (if available) from clinical laboratory assessments performed during the treatment period will be used for the study analysis.
- After completion of the last follow-up visit at 12 weeks following chemotherapy in the first 10
  participants, the Data Monitoring Committee (DMC) will conduct a visual assessment of the
  scans and provide recommendations for the continuation or termination of the Phase II study.






Version: 021 Page: **23 of 96** 

The following table summarizes all the procedures and evaluations to be conducted during the study:

| Study Procedures | First UOHI Evaluation (Screening within 2 weeks prior to the start of AC treatment) | Second UOHI Evaluation (After the 2 <sup>nd</sup> cycle of doxorubicin and before te 3 <sup>rd</sup> cycle) | Third UOHI Evaluation (After the 4th cycle of doxorubicin and within 2 weeks) | Fourth UOHI<br>Evaluation (12<br>weeks after the<br>4 <sup>th</sup> cycle of<br>doxorubicin) |
|---|---|---|---|---|
| Written informed consent | X | | | |
| Inclusion/exclusion criteria | Х | | | |
| Medical history/review | Х | Х | Х | Х |
| Concomitant medications | Х | Х | Х | Х |
| Height <sup>1</sup> , weight, BMI | Х | Х | Х | Х |
| Vital signs (BP, HR) | Х | Х | Х | Х |
| Lab analysis <sup>2</sup> | Х | | | Х |
| Immunogenicity by ELISA <sup>3</sup> | Х | | | Х |
| Cardiotoxicity biomarkers (troponin and BNP) | Х | Х | Х | Х |
| Pregnancy test | Х | Х | Х | Х |
| Cardiac Magnetic Resonance Imaging | Х | Х | Х | Х |
| rhAnnexin V-128<br>administration and<br>SPECT/CT and Planar<br>imaging | Х | Х | Х | Х |
| Adverse Events | X | X | Х | Х |

<sup>&</sup>lt;sup>1</sup> The height will only be measured at screening.

#### 4.3.5 Planned sample size

Sample size was estimated for the comparison of  $^{99m}$ Tc-rhAnnexin V-128 uptake in doxorubicin treated patients imaged after 2 cycles of doxorubicin versus normal baseline uptake using a 5% significance level and power of 95%. The measured heart uptake in 6 normal females (age 29.5 ± 4.6 years, mean ± SD) was 1.2 ± 0.2% ID/g in the phase I study. Sample size estimations were done

<sup>&</sup>lt;sup>2</sup> See Section 4.3.3.3.2. Additionally, results from laboratory analysis conducted during the oncology treatment will be used for research analysis.

<sup>&</sup>lt;sup>3</sup> Anti-rhAnnexin V-128 IgG and IgM antibodies will be quantified in serum samples by ELISA. For this purpose, 10 mL blood samples will be collected at screening and 12 weeks after the last dose of 4 cycles of doxorubicin (before <sup>99m</sup>Tc-rhAnnexin V-128 administration). Serum will be prepared, divided into six aliquots and frozen (-80°C). Three out of six serum samples per time-point will be shipped to the central laboratory




Version: 021 Page: **24 of 96** 

assuming results in the baseline studies of the patients will be similar to the normal females in the phase I study.

For the comparison of <sup>99m</sup>Tc-rhAnnexin V-128 uptake using a paired analysis and assuming a similar SD of 0.2%, a sample size of 26 patients will allow to detect a change of 0.15 %ID/g with a two-sided 5% significance level and a power of 95% (difference between two dependent means).

For the comparison of left ventricular ejection fraction (LVEF) measured with CMR, a sample size of 28 patients will detect an absolute difference of 5% LVEF units with a two-sided 5% significance level and a power of 95% using a paired analysis and assuming a SD of 7 (difference between two dependent means). Assumptions were based on representative CMR data for LVEF of  $58 \pm 7\%$  from 53 participants with breast cancer, lymphoma, leukemia and myelodysplastic syndrome.

The final study population for recruitment size will be 30 patients, allowing for 5 to 10% patient attrition or incomplete imaging data.




Version: 021 Page: **25 of 96** 

#### 5 SUBJECT POPULATIONS (ANALYSIS SETS)

#### 5.1 Efficacy

#### 5.1.1 Full analysis set (FAS)

In accordance with the Intention To Treat (ITT) principle the FAS population includes all subjects who received the study drug and completed at least one <sup>99m</sup>Tc-rhAnnexin V-128 imaging procedure.

#### 5.1.2 Per Protocol population (PP)

All subjects in the FAS population for whom no major protocol violations/deviations occurred and have attended all the scheduled visits. The criteria defining the major protocol deviations will be established before the data base locking.

#### 5.2 Safety set

The safety population is made up of all subjects who received at least one administration of <sup>99m</sup>Tc-rhAnnexin V-128.

#### 5.3 Primary population

The primary and secondary efficacy analysis will be based on the FAS population.

The assessment of safety and tolerability will be based on the Safety population.




Version: 021 Page: **26 of 96** 

#### **6 STATISTICAL METHODS**

#### 6.1 Statistical analysis strategy

The statistical analyses will be performed in accordance with the principles of ICH E9 guideline and the guideline on clinical evaluation of diagnostic agents and they will be based on data from the study site, unless otherwise stated.

#### 6.1.1 Efficacy endpoint(s)

#### 6.1.1.1 Primary endpoint of PoC

Image quality, imaging agent uptake and clinical relevance of apoptosis imaging in the evaluation of doxorubicin-induced cardiotoxicity in patients with early stage of breast cancer using <sup>99m</sup>Tc-rhAnnexin V-128 will be determined by the DMC (visual image review and consensus). Parameters used by DMC to assess primary endpoint of PoC will be appended to the CSR.

#### 6.1.1.2 Primary endpoint of Phase II

Given the early discontinuation of the study, and the fact that only 2 patients were enrolled in the Phase II part of the study, the efficacy endpoints of the Phase II will not be addressed. Any efficacy data collected for these 2 patients will be provided in patients data listings in addition to the results from the PoC phase.

#### 6.1.1.3 Secondary endpoints

The secondary efficacy endpoints will not be addressed for the same reason as the primary efficacy endpoint for the Phase II part of the study.

#### 6.1.2 Safety endpoint(s)

Safety and tolerability will be primarily evaluated by the incidence of adverse events, clinical laboratory values (hematology, blood chemistry and urinalysis), development of anti-annexin V-128 antibodies, vital signs (blood pressure and heart rate), and physical examination findings.




Version: 021 Page: **27 of 96** 

All safety data will be included in the data listings and summary tables will be based on the safety population. The statistical analysis of safety data will be mainly descriptive in nature.

For continuous variables, descriptive summary statistics will include the number of non-missing values, number of missing values, mean, standard deviation, 95% 2-sided confidence interval, median, lower and upper quartile, minimum and maximum. Box plot graphs will also be presented when appropriate.

For categorical variables, descriptive summary statistics will include counts and percentages per category. Staked column graphs or pie graphs will also be computed if appropriate.

For analysis purposes, baseline for a given assessment will be defined as the last non-missing value prior to the administration of <sup>99m</sup>Tc-rhAnnexin V-128, unless stated otherwise.

#### 6.1.2.1 Adverse events

All original AE/SAE terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 19.0.

Adverse events (AEs) will be listed on an individual basis, including relationship and severity, PT (Preferred Term) and verbatim term. Treatment Emergent Adverse Events (TEAEs) and Adverse Drug Reactions (ADRs) will be summarized by System Organ Class (SOC) and Preferred Term (PT). Patients with more than one adverse event within a particular SOC and PT will be counted only once for that SOC and PT reporting the highest level in severity. The incidence of TEAEs and ADRs will also be summarized by severity.

Listings and summaries of serious adverse events (SAEs), adverse events leading to withdrawal and listings of deaths will also be presented.

Treatment Emergent Adverse Events and Adverse Drug Reactions will be defined as below:

- Treatment Emergent Adverse Events: Events that emerge after the first <sup>99m</sup>Tc-rhAnnexin V-128 injection and up to 30 days after the last injection that were absent before it or worsen relative to the pre-treatment state.
- Adverse Drug Reactions: Treatment emergent adverse events possibly or probably related to study treatment.

#### 6.1.2.2 Clinical laboratory values

Hematology and blood chemistry values are recorded at each imaging visit (4 visits) while urinalysis and immunogenicity values are recorded only at baseline, for screening, and after 12 weeks of the




Version: 021 Page: **28 of 96** 

last cycle of doxorubicin. Patients data listings of all laboratory data collected during the study will be provided. Any abnormal results (both clinically and non-clinically relevant) will also be flagged in the listings.

#### 6.1.2.3 Vital signs and medical review

Medical review data are recorded once at each imaging visit (4 visits) while vital signs data are recorded twice at each imaging visit (4 visits), before the injection of <sup>99m</sup>Tc-rhAnnexin V-128 and at the end of last SPECT/CT procedure (within 2 hrs after <sup>99m</sup>Tc-rhAnnexin V-128 injection). Patients data listings of all vital signs collected during the study will be provided.

#### 6.1.3 Missing data and outliers

#### 6.1.3.1 Missing data

As stated in the protocol, missing data will not be replaced.

#### 6.1.3.2 Missing or incomplete dates

Incomplete dates due to missing day will be recorded as full dates replacing the missing day with the first day of month (01). Incomplete dates due to missing day and month will be recorded as full dates replacing the missing day and month with the first day of month and first month of the year (01/January). The trial database will record the information about incomplete dates due to missing day or due to missing day and month.

Only the incomplete dates related to medical history (date of diagnosis and end date), concomitant medications (start and end date) and AEs (start and end date) will be replaced according to the above rule.

Calculation, sorting or assignation based on dates, in case of incomplete dates, will be performed using the related full dates defined by the above rule.

In all listings, missing dates will be missing and incomplete dates will be reported as full dates. In all listings will also be reported the information about incomplete dates according to the following coding: missing value = full date, Day = missing day, Day&Month = missing day and month.




Version: 021 

#### 6.1.3.3 **Outliers**

For categorical or score data, like adverse events, physical exam's findings and disease assessment parameters, outliers are not expected.

Demographic, vital signs, and clinical laboratory (hematology, blood chemistry and urinalysis) parameters will be checked for outliers according to data plausibility, normal ranges and the range between ± 2 S.D.

For each identified outlier, will inform the Sponsor in order to assess any errors. If data cannot be verified or if relevant, the descriptive statistics of the related parameters will be reported with and without the outliers. If appropriate, outliers can also be specifically identified in the boxplots.

#### 6.1.4 Subject disposition

A listing of dates of assessments (relative day) and their study exposure will be presented by subject.

A summary table and a flow chart will be presented for each subject population presenting the number of subjects at each assessment procedure and identifying the number of subjects who withdrew over time.

#### 6.1.5 Withdrawals

Discontinued subjects will be listed and a summary table of the number and percentage of subjects who withdrew from the study and the reasons for withdrawal will be presented for all screened subjects.

#### 6.1.6 Demographic and baseline characteristics

All demographic and baseline characteristics will be listed by subject. Summary statistics will be provided for demographic and baseline characteristics for FAS population.

#### 6.1.7 Medical and surgical history

Medical and surgical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 19.0.

Medical and surgical history will be listed on an individual basis, including Preferred Term (PT) and verbatim term; the listings will be sorted by subject.




Version: 021 Page: **30 of 96** 

#### 6.1.8 Subject compliance

After reconstitution and radiolabeling, <sup>99m</sup>Tc-rhAnnexin V-128 is administered as a single intravenous bolus of 350 MBq ± 10% at each imaging visit (4 visits). The administered dose recorded in the eCRF will not be the difference between the pre-injection dose and the post-injection residual dose but will be the decay corrected dose which takes into account the natural product half-life.

A listing will be presented for imaging product administration (dose, quality, date) by subject. Deviations from observed and scheduled times will be presented. Summary tables will be presented for all the continuous variables.

A listing will be presented for important concomitant medications.

All the protocol deviations will be also listed by subject.

#### 6.1.9 Prior and concomitant therapies

Concomitant therapies will be coded using ATC Drug Dictionary Version 2016.

Listings will be presented for ATC name (third level) and verbatim text. The listings will be sorted by subject, chronological start date, ATC name, verbatim text and active substance.

#### 6.1.10 Derived data

The derived data are variables which are calculated from the raw data in the eCRF and not included in the database (e.g.: Age, BMI). The formula used for derived data and the strategy for missing data are provided in Section 12.1.

#### 6.1.11 Visit windows

The screening visit (Screening Visit Part 1) can occur anytime within 2 weeks before the injection day (Screening Visit Part 2 – First IP injection and CMRI).

The first follow-up visit (Visit 2) should occur within 24 to 48 hrs after 2<sup>nd</sup> doxorubicin cycle. The second follow-up visit (Visit 3) should occur within 24 to 48 hrs after 4<sup>th</sup> doxorubicin cycle. The third and last follow-up visit (Visit 4) should occur 12 weeks after 4<sup>th</sup> doxorubicin cycle.

#### 6.1.12 Rules and data formats

Data will be presented using an appropriate number of decimal places (i.e. the number of decimal places used does not imply undue precision). Raw data will be presented to the number of decimal places collected, and derived data will be presented to an appropriate number of decimal places.




Version: 021 Page: **31 of 96** 

The appropriate number of decimal places will be determined by general practice, mathematical rationale or scientific rationale (e.g. age should be presented in whole numbers).

For summary statistics, the following will be presented: number of non-missing values (n), number of missing values, arithmetic mean, standard deviation, median, the IQR (first quartile, third quartile), the range (minimum, maximum) and, only if appropriate, 95% 2-sided confidence interval.

Mean, standard deviation, first quartile, median, third quartile and confidence interval values will be rounded to one more decimal place than the raw data whereas minimum and maximum will be reported with the same precision as the raw data.

Percentages will be reported to one decimal place. Percentages will be calculated using a denominator of all subjects in a specified population. The denominator will be specified in a footnote to the tables for clarification if necessary.

p-values will be reported to four decimal places (e.g.: p=0.0037), after rounding; p-values which are less than 0.0001 will be presented as "<0.0001".

All text fields must be left justified and numeric or numeric with some text specification (e.g. not done, unknown, <4.5, ...) must be decimal justified. Dates will be presented in the format [dd/mm/yyyy] and times in the format [hh:mm] using 24-hour clock scale.

#### 6.1.13 Pooling of centres

Not applicable.

#### 6.1.14 Interim analysis

No formal interim analysis will be done; however the DMC will review the images of the first 10 participants of the study to determine the feasibility of imaging apoptotic activity in the evaluation of doxorubicin-induced cardiotoxicity.

## 6.1.15 Role of independent data monitoring committee (DMC) / interim data review committee

The Data Monitoring Committee (DMC) consists of investigators and Sponsor representatives, as well as external persons such as independent experts, if deemed necessary by the Sponsor. The main function of the committee will be to review and evaluate the images of the first 10 participants in terms of image quality, visual efficacy (uptake) and clinical relevance of the study product, and determine if there is a significant evidence of inadequate technical performance in this study group. The DMC will also determine if there is an excess of adverse events.




Version: 021 Page: **32 of 96** 

The DMC will promptly give recommendations to continue or terminate the study. The DMC report will be prepared by the Sponsor and sent to the REB and regulatory authorities as required. Preliminary results can be used by the Sponsor for publication purpose, before the end of the main trial.

#### 6.1.16 Covariates and analysis of subgroups

Not applicable.

#### 6.1.17 Sensitivity analysis

Not applicable.

#### 6.1.18 Multiplicity

As stated in the protocol, no adjustements will be made for multiplicity.

#### 6.1.19 Significance testing and estimation

Not applicable.




Version: 021 Page: **33 of 96** 

# 7 COMPUTER SYSTEMS, SOFTWARE AND VALIDATION OF PROGRAMS

#### 7.1 Hardware

The statistical analysis will be performed using Dell personal computer with Windows 7 professional (64 bit) as operating system.

#### 7.2 Software

All tables, listings and figures will be produced and statistical analysis performed using SAS version 9.4. All output will be in Word format.

#### 7.3 Validation programs

An Independent Statistician is responsible for reviewing each project program and output associated with the deliverable product. Program logs are reviewed for logical, syntax and fatal errors. The review in SAS includes, but is not limited to, all ERRORS, WARNINGS, NOTES, and variables check. Program logs are also reviewed for accurate and consistent variable and observation counts following each procedure and data step.

The Independent Statistician is also responsible for checking and reviewing the work produced using whatever method he/she feels is appropriate (e.g. SAS commands review, hand calculation, etc.) to reassure of the quality of the output.

Outputs are reviewed for typographical errors, misspellings and nonsensical values or results and to check the consistency with the reporting and analysis plan. Outputs are cross-checked against each other for accuracy and consistency. For statistical tables, listings, and figures, this procedure includes comparison of subject group numbers, counts of subjects at each observation point, and consistency of results for variables between outputs.

Findings of the quality control reviews are communicated to the party responsible for making necessary changes. The programs will be retested after modifications.

After final review, and when no further changes are required to produce the deliverable, the Independent Statistician needs to complete and sign the SAS Outputs, to indicate that he has successfully performed all of his responsibilities.


Version: 021 Page: **34 of 96** 

#### 8 CHANGES FROM PROTOCOL

As per the sponsor decision, it was decided to close the study after the first 12 patients were enrolled. For this reason and due to the small number of patients included in the protocol, the efficacy analyses will be reduced to the analyses presented during the proof of concept meeting (10 patients) and the imaging data from the 2 additional patients will be presented in subjects data listings. In addition, summaries of demography, subject disposition and adverse events will be provided and any additional data will be presented in subjects data listings and the results described in a short close-out CSR.




Version: 021 Page: **35 of 96** 

### 9 REFERENCES

Not applicable.




Version: 021 Page: **36 of 96** 

#### 10 DATA PRESENTATION

Data listings are presented for all screened subjects.

Footnotes should be used to clarify ambiguities (e.g.: the denominator used to calculate a percentage or notes for the programmer). If the number of footnotes is high, they could be presented only in the last page, with on each page the following footnote "See last page for listing notes". The order of the footnotes for key symbols (\*, ~) will be in the order that they appear in the listing.

#### 10.1 Listings index

#### **16.2 SUBJECT DATA LISTINGS**

#### 16.2.1 Discontinued subjects

Listing 16.2.1.1: Subject Disposition – All Subjects

Listing 16.2.1.2: Subject Disposition – Study Withdrawals

Listing 16.2.1.3: Inclusion Criteria

Listing 16.2.1.4: Exclusion Criteria

Listing 16.2.1.5: Screening Failures

#### 16.2.2 Protocol deviations

Listing 16.2.2: Protocol Deviations and Reasons for Exclusion from the Study

**Populations** 

#### 16.2.3 Subjects excluded from the efficacy analysis

Not applicable

#### 16.2.4 Demographic data

Listing 16.2.4.1: Demographics

Listing 16.2.4.2: Medical History and Associated Pathologies

Listing 16.2.4.3: Prior and Concomitant Medications

#### 16.2.5 Compliance and/or drug concentration data

Listing 16.2.5.1: Study Drug Administration and Extent of Subject Exposure

Listing 16.2.5.2: Chemotherapy Treatment

#### 16.2.6 Individual efficacy response data

Listing 16.2.6.1: Imaging Assessment

Listing 16.2.6.2: Cardiac Magnetic Resonance Imaging


Version: 021 Page: **37 of 96** 

Listing 16.2.6.3: Cardiotoxicity Biomarkers

#### 16.2.7 Adverse event listings (each subject)

Listing 16.2.7.1: All Adverse Events

Listing 16.2.7.2: Serious Adverse Events

Listing 16.2.7.3: Adverse Events Leading to Withdrawal

Listing 16.2.7.4: Adverse Events with Outcome Death

#### 16.2.8 Listing of individual laboratory measurements by subject

Listing 16.2.8.1: Hematology

Listing 16.2.8.2: Blood Chemistry

Listing 16.2.8.3: Urinalysis

Listing 16.2.8.4: Immunogenicity

#### 16.2.9 Listing of other safety data

Listing 16.2.9.1: Pregnancy Test

Listing 16.2.9.2: Pregnancy Test (Before CMRI Procedure)

Listing 16.2.9.3: Medical Review

Listing 16.2.9.4: Vital Signs

### 10.2 Listing templates

Listing templates are provided in Appendix 11.1. The listings will be presented in landscape, in a fixed font (Arial) with a minimum size as 8.

#### 10.3 Tables index

#### 14. TABLES, FIGURES AND GRAPHS

#### 14.1 DEMOGRAPHIC DATA

Table 14.1.1: Subject Disposition

Table 14.1.2: Analysis Populations

Table 14.1.3: Protocol Deviations

Table 14.1.4.1: Demographics – FAS Population

Table 14.1.4.2: Demographics – Safety Population

Table 14.1.5.1: Medical History and Associated Pathologies – Safety Population

| _ | ٠. | | |
|-----|------|---|------|
| ۷,۷ | nfic | n | tio |
| | | | 1111 |

Number (%) of Subjects Reporting Serious Adverse Drug Reactions

|---|---|---|
| | | Version: 021 Page: <b>38 of 96</b> |
| Table | 14.1.6.1: | Prior Medications or Non-Drug Therapies – Safety Population |
| Table | 14.1.6.2: | Prior and Concomitant Medications or Non-Drug Therapies – Safety |
| | | Population |
| Table | 14.1.7.1: | Study Drug Administration – FAS Population |
| Table | 14.1.7.2: | Study Drug Administration – Safety Population |
| Table | 14.1.8.1: | Chemotherapy Treatment – FAS Population |
| Table | 14.1.8.2: | Chemotherapy Treatment – Safety Population |
| 14.2 EFFICACY | DATA | |
| Table | 14.2.1.1: | Primary Efficacy Endpoint – AU (%ID/g) – FAS Population |
| Table | 14.2.1.2: | Primary Efficacy Endpoint – AU (%ID/g) – PP Population |
| Table | 14.2.2.1: | Secondary Efficacy Endpoint – SUV – FAS Population |
| Table | 14.2.2.2: | Secondary Efficacy Endpoint – CUR1 – FAS Population |
| Table | 14.2.2.3: | Secondary Efficacy Endpoint – CUR2 – FAS Population |
| Table | 14.2.2.4: | Secondary Efficacy Endpoint – Cardiac MRI – FAS Population |
| Table | 14.2.3.1: | Cardiotoxicity Biomarkers – FAS Population |
| 14.3 SAFETY D | ATA | |
| 14.3.1 Displays | of Adverse | Events |
| Table | 14.3.1.1: | Overall Summary of Adverse Events – Safety Population |
| Table | 14.3.1.2: | Number (%) of Subjects Reporting Treatment Emergent Adverse |
| | | Events by Primary System Organ Class and Preferred Term - |
| | | Safety Population |
| Table | 14.3.1.3: | Number (%) of Subjects Reporting Treatment Emergent Adverse |
| | | Events by Severity – Safety Population |
| Table | 14.3.1.4: | Number (%) of Subjects Reporting Adverse Drug Reactions by Severity – Safety Population |
| Table | 14.3.1.5: | Number (%) of Subjects Reporting Treatment Emergent Serious |
| | | Adverse Events by Primary System Organ Class and Preferred |
| | | Term – Safety Population |
| Table | 14.3.1.6: | Number (%) of Subjects Reporting Treatment Emergent Serious |
| | | Adverse Events by Severity – Safety Population |

by Severity - Safety Population

Table 14.3.1.7:




Version: 021 Page: **39 of 96** 

#### 14.3.2 Listings of Deaths, Other Serious and Significant Adverse Events

Table 14.3.2.1: Listing of Adverse Events with Outcome Death – Safety Population

Table 14.3.2.2: Listing of Serious Adverse Events – Safety Population

#### 14.3.3 Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events

Only raw narratives will be presented in this section if any.

### 14.3.4 Abnormal Laboratory Value Listing (each patient)

Only patients with clinically significant abnormal laboratory value(s) will be presented in this section if any.

Table 14.3.4: Abnormal Laboratory Value Listing (Each Patient) – Safety Population

#### 14.3.5 Laboratory Measurements

Table 14.3.5.1: Hematology – Safety Population

Table 14.3.5.2: Blood Chemistry – Safety Population

Table 14.3.5.3: Urinalysis – Safety Population

Table 14.3.5.4: Immunogenicity – Safety Population

#### 14.3.6 Other Safety Data

Table 14.3.6.1: Medical Review – Safety Population

Table 14.3.6.2: Vital Signs – Safety Population

### 10.4 Table templates

Table templates are provided for each unique table in Appendix 11.2. The tables will be presented in landscape, in a fixed font (arial) with a minimum size as 8.

All tables, in table number order, must be presented in a single Word file.

### 10.5 Figures index

#### 14. TABLES, FIGURES AND GRAPHS

#### 14.2 EFFICACY DATA

Figure 14.2.1.1: Cardiotoxicity Biomarkers – FAS Population

Figure 14.2.1.1: Primary Efficacy Endpoint – AU (%ID/g) – FAS Population

Figure 14.2.1.2: Primary Efficacy Endpoint – AU (%ID/g) – PP Population




| Figure 14.2.2.1: | Secondary Efficacy Endpoint – SUV – FAS Population |
|---|---|
| Figure 14.2.2.2: | Secondary Efficacy Endpoint – CUR1 – FAS Population |
| Figure 14.2.2.3: | Secondary Efficacy Endpoint – CUR2 – FAS Population |
| Figure 14.2.2.4: | Secondary Efficacy Endpoint – Cardiac MRI – FAS Population |
| Figure 14.2.2.5: | Secondary Efficacy Endpoint – Correlation between Myocardial Uptake and Cardiac MRI – FAS Population |
| Figure 14.2.2.5: | Secondary Efficacy Endpoint – Correlation between Myocardial |
| | Uptake and Cardiotoxicity Biomarkers – FAS Population |
| Figure 14.2.3.1: | Cardiotoxicity Biomarkers – FAS Population |

#### **14.3 SAFETY DATA**

#### 14.3.5 Laboratory Measurements

Figure 14.3.5.1: Hematology – Safety Population

Version: 021

Figure 14.3.5.2: Blood Chemistry – Safety Population

Figure 14.3.5.3: Urinalysis – Safety Population

#### 14.3.6 Other Safety Data

Figure 14.3.6.1: Medical Review – Safety Population

Figure 14.3.6.2: Vital Signs – Safety Population

### 10.6 Figure templates

Figure templates are provided for each unique figure in Appendix 0. The figures will be presented in landscape, in a fixed font (arial) with a minimum size as 8.

All figures, in figure number order, must be presented in a single Word file.

# 10.7 Statistical appendix

A Statistical Appendix for inclusion in the study report will be provided. All the methods used in checking the assumptions of the analyses and conclusions should be included and explained. Transformation of the data or other methods used for the statistical analysis other than the ones detailed in the SAP will be described and the change will be justified. All the SAS output will be included without reworking the data (raw output).




Version: 021 Page: **41 of 96** 

This output should contain the study number, the date, the number of pages printed by SAS and the table number to which it refers. Any other relevant information (e.g. statistical references...) will be added in the statistical appendix.


Version: 021 Page: **42 of 96** 

## 11 APPENDICES

# 11.1 Standard listings

All listings must contain examples of possible data and be presented in fixed font (arial) with a minimum size as 8.




Version: 021 Page: **43 of 96** 

### **Listing 16.2.1.1:** Subject Disposition – All subjects

| | | | | | | | Premature study | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Informed consent date | Screening part 1 date | Screening part 2 date | Visit 2 date | Visit 3 date | Visit 4 date | discontinuation date | FAS | PP | Safety | |
| PAT_PATNUMBER | PAT_INFCONS_DATE | PAT_FIRSTVISITDAT<br>E | PATV_VISITDATE | PATV_VISITDATE | PATV_VISITDATE | PATV_VISITDATE | SD_DATE | [Derived data] | [Derived data] | [Derived data] | - |
| 05-CA-001 | 11/03/2011 | 11/03/2011 | 11/03/2011 | 11/04/2011 | 12/04/2011 | 11/05/2011 | | Yes | Yes | Yes | |
| 05-CA-002 | 09/04/2011 | 09/04/2011 | 09/04/2011 | 09/04/2011 | 10/04/2011 | 10/05/2011 | | Yes | Yes | Yes | |
| 05-CA-003 | 10/07/2011 | 10/07/2011 | 10/07/2011 | 15/07/2011 | 16/07/2011 | NA | 10/08/2011 | Yes | No | Yes | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_SD.

Note: NA = Not Available for patient early withdrawal




Version: 021 Page: **44 of 96** 

## **Listing 16.2.1.2:** Subject Disposition – Study Withdrawals

| | | | Premature study | Reason for | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Informed consent date | Screening part 1 date | discontinuation date | withdrawal | Explanation | Notes | FAS | PP | Safety |
| PAT_PATNUMBER | PAT_INFCONS_DATE | PAT_FIRSTVISITDATE | SD_DATE | SD_OUTCOME | SD_OUTCOME_SP | SD_NOTES | [Derived data] | [Derived data] | [Derived data] |
| 05-CA-001 | 11/03/2011 | 11/03/2011 | 10/05/2012 | XXXXXX | XXXXXX | XXXXXX | Yes | No | Yes |
| 05-CA-002 | 09/04/2011 | 09/04/2011 | 10/05/2012 | XXXXXX | XXXXXX | XXXXXX | Yes | No | Yes |
| 05-CA-003 | 10/07/2011 | 10/07/2011 | 10/05/2012 | XXXXXX | XXXXXX | XXXXXX | Yes | No | Yes |

Data Source Table: W\_PATIENT, W\_SD.

Note: NA = Not Available for patient early withdrawal




Version: 021 Page: **45 of 96** 

## **Listing 16.2.1.3: Inclusion Criteria**

| | | | | Inclusion criteria | |
|---|---|---|---|---|---|
| Subject ID | Age | Screening part 1 date | First | Second | Third |
| PAT_PATNUMBER | PAT_AGEYEAR | PAT_FIRSTVISITDATE | IC_1 | IC_2 | IC_3 |
| 05-CA-001 | 54 | 11/03/2011 | Yes | Yes | No |
| 05-CA-002 | 68 | 09/04/2011 | Yes | Yes | Yes |
| 05-CA-003 | 59 | 10/07/2011 | No | Yes | Yes |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_IEC.

Note: NA = Not Available




Version: 021 Page: **46 of 96** 

## Listing 16.2.1.4: Exclusion Criteria

#### Exclusion criteria

| Subject ID | Age | Screening part 1 date | First | Second | Third | Fourth | Fifth | Sixth | Seventh | Eighth | Ninth | Tenth |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_AGEYEAR | PAT_FIRSTVISITDATE | EC_1 | EC_2 | EC_3 | EC_4 | EC_5 | EC_6 | EC_7 | EC_8 | EC_9 | EC_10 |
| 05-CA-001 | 54 | 11/03/2011 | No | No | No | No | No | No | No | No | No | No |
| 05-CA-002 | 68 | 09/04/2011 | No | Yes | No | No | No | No | No | No | No | No |
| 05-CA-003 | 59 | 10/07/2011 | Yes | No | No | No | No | No | No | No | No | No |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_IEC.

Note: NA = Not Available




Version: 021 Page: **47 of 96** 

## **Listing 16.2.1.5:** Screening Failures

| Subject ID | Screening failure | Reason for screen failure |
|---------------|-------------------|---------------------------|
| PAT_PATNUMBER | [Derived data] | [Derived data] |
| 05-CA-001 | Yes | XXXXX |
| 05-CA-002 | No | XXXXX |
| 05-CA-003 | No | XXXXX |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_IEC, W\_SD.

Note: NA = Not Available




Version: 021 Page: **48 of 96** 

# Listing 16.2.2: Protocol Deviations and Reasons for Exclusion from the Study Populations

| Subject ID | Screening part 1 date | FAS | PP | Safety | Deviation description | Reason for exclusion |
|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_FIRSTVISITDATE | [Derived data] | [Derived data] | [Derived data] | [Derived data] | [Derived data] |
| 05-CA-001 | 11/03/2011 | Yes | Yes | No | XXXXXX | XXXXXX |
| 05-CA-002 | 09/04/2011 | No | Yes | Yes | XXXXXX | XXXXXX |
| 05-CA-003 | 10/07/2011 | Yes | No | Yes | XXXXXX | XXXXXX |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_SD.

Note: NA = Not Available




Version: 021 Page: **49 of 96** 

# Listing 16.2.4.1: Demographics

| Subject ID | Screening part 1 date | Date of birth (month/year) | Age | Ethnicity | Specify other ethnicity |
|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_FIRSTVISITDATE | PAT_BIRTH_MONTH<br>PAT_BIRTH_YEAR | PAT_AGEYEAR | PAT_ETHNIC | PAT_ETHNIC_SP |
| 05-CA-001 | 11/03/2011 | 03/1959 | 54 | Other | XXXXXXX |
| 05-CA-002 | 09/04/2011 | 09/1945 | 68 | Caucasian | |
| 05-CA-003 | 10/07/2011 | 02/1954 | 59 | Asian | |




Version: 021 Page: **50 of 96** 

## **Listing 16.2.4.2:** Medical History and Associated Pathologies

| Subject ID | Medical condition | Preferred term | Date of diagnosis | Partial date | Ongoing? | Currently treated? | Resolution date | Partial date |
|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | MH_MEDCOND | MEDDRA_PT | MH_DIAGN_DATE | MH_PARTIAL_START<br>_DATE | MH_ONGOING_YN | MH_TREATED_YN | MH_END_DATE | MH_PARTIAL_END_D<br>ATE |
| 05-CA-001 | XXXXXX | XXXXXX | 15/08/1990 | Day | No | | 14/04/1994 | |
| 05-CA-002 | XXXXXX | XXXXXX | 31/12/2007 | | No | | 15/06/2008 | Day&Month |
| 05-CA-003 | XXXXXX | XXXXXX | 05/05/2005 | | Yes | Yes | | |

Data Source Table: W\_PATIENT, W\_MH.

Dictionary Name: MedDRA Version: 19.0

Note: NA = Not Available




Version: 021 Page: **51 of 96** 

## **Listing 16.2.4.3/1: Prior and Concomitant Medications**

| | Medication | ATC description | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | trade name | (third level) | Enrollment date | Start date (day) | Partial date | Ongoing? | End date | Partial date |
| PAT_PATNUMBER | CM_NAME | ATC_LV3_DESCR | PAT_FIRSTVISITDATE | CM_START_DATE | CM_PARTIAL_START_<br>DATE | CM_ONGOING_YN | CM_END_DATE | CM_PARTIAL_END_D<br>ATE |
| 05-CA-001 | XXXXXXX | XXXXXX | 11/03/2011 | 15/08/1990 (xx) | Day | No | 14/04/1994 | Day |
| 05-CA-002 | XXXXXXX | XXXXXX | 09/04/2011 | 31/12/2007 (xx) | Day&Month | No | 15/06/2008 | Day&Month |
| 05-CA-003 | XXXXXXX | XXXXXX | 10/07/2011 | 05/05/2005 (xx) | | Yes | | |

Data Source Table: W\_PATIENT, W\_CM.

Dictionary Name: ATC Version: 2016

Note: NA = Not Available




Version: 021 Page: **52 of 96** 

## **Listing 16.2.4.3/2: Prior and Concomitant Medications**

| | Medication | ATC description | | | | Frequency of | | Route of | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | trade name | (third level) | Total daily dose | Unit | Specify other unit | administration | Specify other frequency | administration | Specify other route |
| PAT_PATNUMBER | CM_NAME | ATC_LV3_DESCR | CM_DOSE | CM_DOSEU | CM_DOSEU_SP | CM_FREQ | CM_FREQ_SP | CM_ROUTE | CM_ROUTE_SP |
| 05-CA-001 | XXXXXXXX | XXXXXX | 3 | G | | BID | | Otherl | XXXXXX |
| 05-CA-002 | XXXXXXXX | XXXXXX | 3 | Other | XXXXXX | TID | | Intramuscolar | |
| 05-CA-003 | XXXXXXX | XXXXXX | 12 | Mg | | Other | XXXXXX | Subcutaneous | |

Data Source Table: W\_PATIENT, W\_CM.

Dictionary Name: ATC Version: 2016

Note: NA = Not Available




Version: 021 Page: **53 of 96** 

## Listing 16.2.5.1/1: Study Drug Administration and Extent of Subject Exposure

| | | | Has the injection | Reason for not | | | | Batch of |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Visit | Visit date | been performed? | performing the injection | Injection date | Injection time | Batch of kit | 99mTc generator |
| PAT_PATNUMBER | VISIT_NAME | PATV_VISITDATE | ANN_YN | ANN_YN_SP | ANN_DATE | ANN_TIME | ANN_KIT | ANN_GEN |
| 05-CA-001 | Screening part 1 | 10/03/2011 | Yes | | 11/03/2011 | 10:50 | 09101-110631 | 09101-110631 |
| 05-CA-002 | Screening part 2 | 08/02/2011 | Yes | | 03/03/2011 | 10:00 | 09101-110981 | 09101-110981 |
| 05-CA-002 | Visit 1 | 08/03/2011 | Yes | | 08/03/2011 | 11:00 | 09101-110981 | 09101-111012 |
| 05-CA-003 | Screening part 2 | 01/04/2011 | No | XXXXXXX | | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_ANN.

Note: NA = Not Available




Version: 021 Page: **54 of 96** 

## Listing 16.2.5.1/2: Study Drug Administration and Extent of Subject Exposure

| | | | Has the injection | | Pre injection total | Post injection residual | Actual dose | Volume of administered |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Visit | Visit date | been performed? | Radiochemical purity | activity-dose in the syringe (MBq) | activity-dose in the syringe (MBq) | injected (MBq) | solution (mL) |
| PAT_PATNUMBER | VISIT_NAME | PATV_VISITDATE | ANN_YN | ANN_TEST1 | ANN_TEST2_PRE | ANN_TEST2_POST | ANN_TEST2_EFF | ANN_TEST2_VOL |
| 05-CA-001 | Screening part 1 | 10/03/2011 | Yes | 98.7% | 123 | 123 | 123 | 123 |
| 05-CA-002 | Screening part 2 | 08/02/2011 | Yes | 99.1% | 456 | 456 | 456 | 456 |
| 05-CA-002 | Visit 1 | 08/03/2011 | Yes | 99.1% | 789 | 789 | 789 | 789 |
| 05-CA-003 | Screening part 2 | 01/04/2011 | No | | | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_ANN.

Note: NA = Not Available




Version: 021 Page: **55 of 96** 

## **Listing 16.2.5.2: Chemotherapy Treatment**

| | | | | Fire | st cycle | Seco | ond cycle | Thir | d cycle | Four | rth cycle | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Has chemotherapy | Chemotherapy | Doxorubicin | Cyclophosphamide | Doxorubicin | Cyclophosphamide | Doxorubicin | Cyclophosphamide | Doxorubicin | Cyclophosphamide | Number |
| Subject ID | Visit date | been started? | start date | dose (mg/m^2) | dose (mg/m^2) | dose (mg/m^2) | dose (mg/m^2) | dose (mg/m^2) | dose (mg/m^2) | dose (mg/m^2) | dose (mg/m^2) | of cycles |
| PAT_PATN<br>UMBER | PATV_VISI<br>TDATE | CT_YN | CT_DATE | CT_DOX1 | CT_CYC1 | CT_DOX2 | CT_CYC2 | CT_DOX1 | CT_CYC1 | CT_DOX2 | CT_CYC2 | CT_CT_<br>N |
| 05-CA-001 | 10/03/2011 | Yes | 11/03/2011 | 400 | 250 | 514 | 625 | 514 | 625 | 514 | 625 | 4 |
| 05-CA-002 | 08/02/2011 | Yes | 03/03/2011 | 350 | 400 | 654 | 258 | 654 | 258 | 654 | 258 | 4 |
| 05-CA-003 | 01/04/2011 | No | | | | | | | | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_CT.

Note: NA = Not Available




Version: 021 Page: **56 of 96** 

## **Listing 16.2.6.1/1: Imaging Assessment**

| | | | | | Time from IP | Has the imaging | Reason for non | | | Have images been | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Visit | Visit date | Injection date | Imaging procedure | injection (min) | been completed? | completion | Date | Time | received and reviewed? | |
| PAT_PATNUMBE<br>R | VISIT_NAME | PATV_VISITDATE | ANN_DATE | [Derived data] | [Derived data] | SP_YN<br>SPCT_YN | SP_YN_SP<br>SPCT_YN_SP | SP_DATE<br>SPCT_DATE | SP_TIME<br>SPCT_TIME | SP_REV_YN<br>SPCT_REV_YN | - |
| 05-CA-001 | Screening part 2 | 10/03/2011 | 11/03/2011 | SPECT | 60 | Yes | | 11/03/2011 | 10:50 | Yes | |
| 05-CA-001 | Screening part 2 | 10/03/2011 | 11/03/2011 | SPECT/CT | 120 | Yes | | 11/03/2011 | 10:00 | Yes | |
| 05-CA-002 | Visit 1 | 08/03/2011 | 03/03/2011 | SPECT | 60 | No | XXXXXXX | | | | |
| 05-CA-002 | Visit 1 | 08/03/2011 | 03/03/2011 | SPECT/CT | 120 | Yes | | 08/03/2011 | 15:00 | Yes | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_SPECT\_SPECTCT.

Note: NA = Not Available




Version: 021 Page: **57 of 96** 

### **Listing 16.2.6.1/2: Imaging Assessment**

| | | | | | | | | Up | take | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Visit | Visit date | Injection date | Imaging procedure | Time from IP injection (min) | Has the imaging been completed? | AU (%ID/g) | SUV | CUR1 | CUR2 |
| PAT_PATNUMBER | VISIT_NAME | PATV_VISITDATE | ANN_DATE | [Derived data] | [Derived data] | SP_YN<br>SPCT_YN | SP_RESULT<br>_SPCT_RES<br>ULT | SP_SUV<br>SPCT_SUV | SP_CUR1<br>SPCT_CUR1 | SP_CUR2<br>SPCT_CUR2 |
| 05-CA-001 | Screening part 2 | 10/03/2011 | 11/03/2011 | SPECT | 60 | Yes | 49% | 22,78 | 48,99 | 77,00 |
| 05-CA-001 | Screening part 2 | 10/03/2011 | 11/03/2011 | SPECT/CT | 120 | Yes | 97% | 35,28 | 07,31 | 64,69 |
| 05-CA-002 | Visit 1 | 08/03/2011 | 03/03/2011 | SPECT | 60 | No | | | | |
| 05-CA-002 | Visit 1 | 08/03/2011 | 03/03/2011 | SPECT/CT | 120 | Yes | 98% | 51,28 | 45,13 | 64,29 |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_SPECT\_SPECTCT.

Note: NA = Not Available; AU = Absolute Uptake, SUV = Standardized Uptake Value; CUR = Cardiac Uptake Ratio




Version: 021 Page: **58 of 96** 

## **Listing 16.2.6.2: Cardiac Magnetic Resonance Imaging**

| | | | Has CMRI | Reason for non | | | | Any clinically | First | Second | Third |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Visit | Visit date | been done? | performance | CMRI date | CMRI time | LVEF (%) | relevant finding? | finding | finding | finding |
| PAT_PATNUMBER | VISIT_NAME | PATV_VISITDATE | CMRI_YN | CMRI_YN_SP | CMRI_DATE | CMRI_TIME | CMRI_LVEF | CMRI_REL_YN | CMRI_REL1 | CMRI_REL2 | CMRI_REL3 |
| 05-CA-001 | Screening part 2 | 10/03/2011 | Yes | | 11/03/2011 | 10:50 | 68.5 | No | | | |
| 05-CA-002 | Screening part 2 | 08/02/2011 | Yes | | 03/03/2011 | 10:00 | 72.3 | No | | | |
| 05-CA-003 | Visit 1 | 08/03/2011 | No | XXXXXX | | | 85.9 | Yes | XXXXXXX | XXXXXX | XXXXXX |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_CMRI.

Note: NA = Not Available




Version: 021 Page: **59 of 96** 

## **Listing 16.2.6.3: Cardiotoxicity Biomarkers**

| | | | | | | | Troponir | (µg/L) | NT-proBN | P (ng/L) |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Visit | Visit date | Have blood tests been done? | Reason for non performance | Sample date | Sample time | Not done | Result | Not done | Result |
| PAT_PATNUMBER | VISIT_NAME | PATV_VISITDATE | CB_YN | CB_YN_SP | CB_DATE | CB_TIME | CB_TRO_ND | CB_TRO | CB_NTP_ND | CB_NTP |
| 05-CA-001 | Screening part 2 | 10/03/2011 | Yes | | 11/03/2011 | 10:50 | Yes | | | 68.5 |
| 05-CA-002 | Screening part 2 | 08/02/2011 | Yes | | 03/03/2011 | 10:00 | | 72.3 | Yes | |
| 05-CA-003 | Visit 1 | 08/03/2011 | No | XXXXXXX | | | | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_CB.

Note: NA = Not Available




Version: 021 Page: **60 of 96** 

### Listing 16.2.7.1/1: All Adverse Events

| | | | Primary system | | Study day of | | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Event ID | Event description | organ class | Preferred term | onset (days)§ | Ongoing? | Duration (days) | TEAE <sup>^</sup> |
| PAT_PATNUMBER | ID_WEB | AE_NAME | MEDDRA_SOC | MEDDRA_PT | [Derived data] | AE_ONGOING_YN | [Derived data] | [Derived data] |
| 05-CA-001 | XXX | XXXXXXX | XXXXXX | XXXXXXXX | YY | No | ≥2 | Yes |
| 05-CA-002 | XXX | XXXXXXX | XXXXXX | XXXXXXXX | YY | No | 15 | Yes |
| 05-CA-003 | XXX | XXXXXXX | XXXXXX | XXXXXXXX | YY | Yes | ≥30 | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Dictionary Name: MedDRA Version: 19.0

Note: NA = Not Available

 $<sup>\</sup>S$  Study day of onset is defined as days from first Annexin injection

<sup>^</sup> TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1 File directory: path of directory status from study level downwards /XXXXXX.sas




Version: 021 Page: **61 of 96** 

# Listing 16.2.7.1/2: All Adverse Events

| Subject ID | Event ID | Event description | AE caused premature withdrawal? | SAE | SAE seriousness | Maximal severity | Causal relationship with medication or procedure | Possible cause | Specify other possible cause | TEAE^ | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBE<br>R | ID_WEB | AE_NAME | AE_WITHD_YN | AE_SAE_YN | [Derived data] | AE_MAXSEV | AE_REL | AE_CAUSE | AE_CAUSE_SP | [Derived data] | - |
| 05-CA-001 | XXX | XXXXXXXX | Yes | Yes | XXXXXX / XXXXX | Grade 2 (Moderate) | Possible | Other | XXXXXXXXXX | Yes | |
| 05-CA-002 | XXX | xxxxxxx | No | No | XXXXXX / XXXXX | Grade 1 (Mild) | Unlikely | Pre-existing/<br>underlying<br>disease | xxxxxxxxx | Yes | |
| 05-CA-003 | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 3 (Severe) | Unrelated | Other treatment | XXXXXXXXXX | Yes | |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

^ TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1
File directory: path of directory status from study level downwards /XXXXXX.sas




Version: 021 Page: **62 of 96** 

### Listing 16.2.7.1/3: All Adverse Events

| Subject ID | Event ID | Event description | Action taken | Other action taken | Other action taken, specify | Outcome | TEAE^ |
|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | ID_WEB | AE_NAME | AE_ACT | [Derived data] | AE_ACT_OTH_SP | AE_OUTCOME | [Derived data] |
| 05-CA-001 | XXX | XXXXXXX | No action | XXX/XXXXX/XXX | | Resolved | Yes |
| 05-CA-002 | XXX | XXXXXXX | Dose modification in next<br>treatment | XXX/XXXXX | XXXXXX | Worsened | Yes |
| 05-CA-003 | XXX | XXXXXXX | Unknown | XXX | | Persisting | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

^ TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1




Version: 021 Page: **63 of 96** 

### Listing 16.2.7.2/1: Serious Adverse Events

| | | | Primary system | | | Study day of | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Event ID | Event description | organ class | Preferred term | Lowest level term | onset (days)§ | Ongoing? | Duration (days) | TEAE <sup>^</sup> |
| PAT_PATNUMBER | ID_WEB | AE_NAME | MEDDRA_SOC | MEDDRA_PT | MEDDRA_LLT | [Derived data] | AE_ONGOING_YN | [Derived data] | [Derived data] |
| 05-CA-001 | XXX | XXXXXXX | XXXXXX | XXXXXXX | XXXXXX | YY | No | ≥2 | Yes |
| 05-CA-002 | XXX | XXXXXXX | XXXXXX | XXXXXXX | XXXXXX | YY | No | 15 | Yes |
| 05-CA-003 | XXX | XXXXXXX | XXXXXX | XXXXXXX | XXXXXX | YY | Yes | ≥30 | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Dictionary Name: MedDRA Version: 19.0

Note: NA = Not Available

<sup>§</sup> Study day of onset is defined as days from first Annexin injection

<sup>^</sup> TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1 File directory: path of directory status from study level downwards /XXXXXX.sas




Version: 021 Page: **64 of 96** 

### Listing 16.2.7.2/2: Serious Adverse Events

| Subject ID | Event ID | Event description | AE caused premature withdrawal? | SAE | SAE seriousness | Maximal severity | Causal relationship with medication or procedure | Possible cause | Specify other possible cause | TEAE^ |
|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBE<br>R | ID_WEB | AE_NAME | AE_WITHD_YN | AE_SAE_YN | [Derived data] | AE_MAXSEV | AE_REL | AE_CAUSE | AE_CAUSE_SP | [Derived data] |
| 05-CA-001 | XXX | XXXXXXX | Yes | Yes | XXXXXX / XXXXX | Grade 2 (Moderate) | Possible | Other | XXXXXXXXXX | Yes |
| 05-CA-002 | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 1 (Mild) | Unlikely | Pre-existing/<br>underlying<br>disease | xxxxxxxxx | Yes |
| 05-CA-003 | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 3 (Severe) | Unrelated | Other treatment | XXXXXXXXXX | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

^ TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1 File directory: path of directory status from study level downwards /XXXXXX.sas




Version: 021 Page: **65 of 96** 

### Listing 16.2.7.2/3: Serious Adverse Events

| Subject ID | Event ID | Event description | Action taken | Other action taken | Other action taken, specify | Outcome | TEAE^ |
|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | ID_WEB | AE_NAME | AE_ACT | [Derived data] | AE_ACT_OTH_SP | AE_OUTCOME | [Derived data] |
| 05-CA-001 | XXX | XXXXXXXX | No action | XXX/XXXXX/XXX | | Resolved | Yes |
| 05-CA-002 | XXX | XXXXXXX | Dose modification in next<br>treatment | XXX/XXXXX | XXXXXX | Worsened | Yes |
| 05-CA-003 | XXX | XXXXXXX | Unknown | XXX | | Persisting | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

^ TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1




Version: 021 Page: **66 of 96** 

### Listing 16.2.7.3/1: Adverse Events Leading to Withdrawal

| | | | Primary system | | Study day of | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Event ID | Event description | organ class | Preferred term | onset (days)§ | Ongoing? | Duration (days) | TEAE <sup>^</sup> | _ |
| PAT_PATNUMBER | ID_WEB | AE_NAME | MEDDRA_SOC | MEDDRA_PT | [Derived data] | AE_ONGOING_YN | [Derived data] | [Derived data] | |
| 05-CA-001 | XXX | XXXXXXX | XXXXXX | XXXXXXX | YY | No | ≥2 | Yes | |
| 05-CA-002 | XXX | XXXXXXX | XXXXXX | XXXXXXX | YY | No | 15 | Yes | |
| 05-CA-003 | XXX | XXXXXXX | XXXXXX | XXXXXXX | YY | Yes | ≥30 | Yes | |

Data Source Table: W\_PATIENT, W\_AE.

Dictionary Name: MedDRA Version: 19.0

Note: NA = Not Available

^ TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1
File directory: path of directory status from study level downwards /XXXXXX.sas

 $<sup>\</sup>S$  Study day of onset is defined as days from first Annexin injection




Version: 021 Page: **67 of 96** 

### Listing 16.2.7.3/2: Adverse Events Leading to Withdrawal

| Subject ID | Event ID | Event description | AE caused premature withdrawal? | SAE | SAE seriousness | Maximal severity | Causal relationship with medication or procedure | Possible cause | Specify other possible cause | TEAE^ |
|---|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBE<br>R | ID_WEB | AE_NAME | AE_WITHD_YN | AE_SAE_YN | [Derived data] | AE_MAXSEV | AE_REL | AE_CAUSE | AE_CAUSE_SP | [Derived data] |
| 05-CA-001 | XXX | XXXXXXXX | Yes | Yes | XXXXXX / XXXXX | Grade 2 (Moderate) | Possible | Other | XXXXXXXXXX | Yes |
| 05-CA-002 | XXX | xxxxxxx | No | No | XXXXXX / XXXXX | Grade 1 (Mild) | Unlikely | Pre-existing/<br>underlying<br>disease | XXXXXXXXXX | Yes |
| 05-CA-003 | XXX | XXXXXXX | No | No | XXXXXX / XXXXX | Grade 3 (Severe) | Unrelated | Other treatment | XXXXXXXXXX | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

^ TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1 File directory: path of directory status from study level downwards /XXXXXX.sas




Version: 021 Page: **68 of 96** 

### Listing 16.2.7.3/3: Adverse Events Leading to Withdrawal

| Subject ID | Event ID | Event description | Action taken | Other action taken | Other action taken, specify | Outcome | TEAE^ |
|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | ID_WEB | AE_NAME | AE_ACT | [Derived data] | AE_ACT_OTH_SP | AE_OUTCOME | [Derived data] |
| 05-CA-001 | XXX | XXXXXXX | No action | XXX/XXXXX/XXX | | Resolved | Yes |
| 05-CA-002 | XXX | XXXXXXX | Dose modification in next<br>treatment | XXX/XXXXX | XXXXXX | Worsened | Yes |
| 05-CA-003 | XXX | XXXXXXX | Unknown | XXX | | Persisting | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

^ TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1




Version: 021 Page: **69 of 96** 

### Listing 16.2.7.4/1: Adverse Events with Outcome Death

| | | | Primary system | | Study day of | | |
|---|---|---|---|---|---|---|---|
| Subject ID | Event ID | Event description | organ class | Preferred term | onset (days)§ | Duration (days) | TEAE <sup>^</sup> |
| PAT_PATNUMBER | ID_WEB | AE_NAME | MEDDRA_SOC | MEDDRA_PT | [Derived data] | [Derived data] | [Derived data] |
| 05-CA-001 | XXX | XXXXXXX | XXXXXX | XXXXXXXX | YY | ≥2 | Yes |
| 05-CA-002 | XXX | XXXXXXX | XXXXXX | XXXXXXXX | YY | 15 | Yes |
| 05-CA-003 | XXX | XXXXXXX | XXXXXX | XXXXXXXX | YY | ≥30 | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Dictionary Name: MedDRA Version: 19.0

Note: NA = Not Available

 $<sup>\</sup>S$  Study day of onset is defined as days from first Annexin injection

<sup>^</sup> TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1
File directory: path of directory status from study level downwards /XXXXXX.sas




Version: 021 Page: **70 of 96** 

#### Listing 16.2.7.4/2: Adverse Events with Outcome Death

AE caused premature Specify other Causal relationship with SAE TEAE^ Event ID Subject ID Event description withdrawal? SAE seriousness Maximal severity medication or procedure Possible cause possible cause PAT\_PATNUMBE ID\_WEB AE\_NAME AE\_WITHD\_YN AE\_SAE\_YN AE\_MAXSEV AE\_REL AE\_CAUSE AE\_CAUSE\_SP [Derived data] [Derived data] 05-CA-001 XXX XXXXXXXX Yes XXXXXX / XXXXX Grade 2 (Moderate) XXXXXXXXXX Yes Possible Other Yes Pre-existing/ 05-CA-002 XXXXXXXXXXX No No XXXXXX / XXXXX Grade 1 (Mild) Unlikely underlying XXXXXXXXXX Yes disease Other 05-CA-003 XXX XXXXXXX No No XXXXXX / XXXXX Grade 3 (Severe) Unrelated XXXXXXXXXX Yes treatment

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

^ TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1 File directory: path of directory status from study level downwards /XXXXXX.sas




Version: 021 Page: **71 of 96** 

### Listing 16.2.7.4/3: Adverse Events with Outcome Death

| Subject ID | Event ID | Event description | Action taken | Other action taken | Other action taken, specify | Outcome | TEAE^ |
|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | ID_WEB | AE_NAME | AE_ACT | [Derived data] | AE_ACT_OTH_SP | AE_OUTCOME | [Derived data] |
| 05-CA-001 | XXX | XXXXXXX | No action | XXX/XXXXX/XXX | | Resolved | Yes |
| 05-CA-002 | XXX | XXXXXXX | Dose modification in next treatment | XXX/XXXXX | XXXXXX | Worsened | Yes |
| 05-CA-003 | XXX | XXXXXXX | Unknown | XXX | | Persisting | Yes |

Data Source Table: W\_PATIENT, W\_AE.

Note: NA = Not Available

^ TEAE: Treatment Emegent Adverse Event as defined in paragraph 6.1.2.1




Version: 021 Page: **72 of 96** 

# Listing 16.2.8.1/1: Hematology

| Subject ID | Visit | Have hematology tests been done? | Sample collection date | Sample collection time | Parameter | Result | Unit | Abnormality |
|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | VISIT_NAME | HE_YN | HE_DATE | HE_TIME | | HE_RBC | | HE_RBC_ABN |
| 05-CA-001 | Screening part 1 | Yes | 11/03/2011 | 10:52 | Red Blood Cells | 99.99 | 10 <sup>12</sup> /L | Abnormal Non-Clinical Relevant |
| | | | | | Hematocrit | 99.99 | L/L | Abnormal Non-Clinical<br>Relevant |
| 05-CA-001 | Visit 2 | Yes | 09/04/2011 | 15:00 | | | | |
| 05-CA-002<br>05-CA-003 | Screening part 1<br>Visit 4 | Yes<br>No: XXXXX | 10/07/2011 | Not done | | | | |



Version: 021 Page: **73 of 96** 

Listing 16.2.8.2/1: Blood Chemistry

Repeat listing 16.2.8.1 for chemistry parameters




Version: 021 Page: **74 of 96** 

Listing 16.2.8.3/1: Urinalysis

Repeat listing 16.2.8.1 for urinalysis parameters




Version: 021 Page: **75 of 96** 

# Listing 16.2.8.4: Immunogenicity

| | | Has venous | Reason for non | | | |
|---|---|---|---|---|---|---|
| <br>Subject ID | Visit | sample been done? | performance | Sample collection date | Sample collection time | Result |
| PAT_PATNUMBER | VISIT_NAME | IM_YN | IM_YN_SP | IM_DATE | IM_TIME | [Provided data] |
| 05-CA-001 | Screening part 1 | Yes | | 11/03/2011 | 10:52 | Negative |
| 05-CA-001 | Visit 4 | Yes | | 09/04/2011 | 15:00 | Positive |
| 05-CA-002 | Screening part 1 | Yes | | 10/07/2011 | 09:38 | Positive |
| 05-CA-003 | Visit 4 | No | XXXXXXXXX | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_IM. Other data source: database provided by Sponsor: XXXXXXXX.

Note: NA = Not Available




Version: 021 Page: **76 of 96** 

# **Listing 16.2.9.1: Pregnancy Test**

| Subject ID | Age | Visit | Has the pregnancy test been performed? | Reason for non performance | Specify reason | Pregnancy<br>test date | Pregnancy<br>test time | Pregnancy<br>test result | _ |
|---|---|---|---|---|---|---|---|---|---|
| PAT_PATNUMBER | PAT_AGEYEAR | VISIT_NAME | PT_YN | PT_NOTDONE | PT_NOTDONE_SP | PT_DATE | PT_TIME | PT_RESULT | • |
| 05-CA-001 | 54 | Screening part 1 | Not applicable | | | | | | |
| 05-CA-001 | 54 | Visit 2 | Not applicable | | | | | | |
| 05-CA-002 | 38 | Screening part 1 | Yes | | | 09/04/2011 | 12:00 | Negative | |
| 05-CA-002 | 38 | Visit 4 | Yes | | | 12/04/2011 | 10:00 | Negative | |
| 05-CA-003 | 59 | Visit 3 | No | Menopause | | | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_PT.

Note: NA = Not Available




Version: 021 Page: **77 of 96** 

# **Listing 16.2.9.3:** Physical Examination

| | | | | | | | | | | | Specify | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Visit | Has the physical examination been done? | Reason for non performance | Physical examination date | Physical examination time | Height (cm) | Weight (Kg) | BMI (Kg/m^2) | Any clinically relevant finding? | First finding | Second finding | Third finding |
| | | | | | | <u> </u> | 0 ( 0/ | | | | | |
| PAT_PATNUMBER | VISIT_NAME | MR_YN | MR_YN_SP | MR_DATE | MR_TIME | HEIGHT | WEIGHT | BMI | MR_RELFIND_YN | MR_RELFIND1 | MR_RELFIND2 | MR_RELFIND3 |
| 05-CA-001 | Screening part | Yes | | 09/04/2011 | 12:00 | 180 | 68.5 | 23.8 | No | | | |
| 05-CA-002 | Visit 2 | No | XXXXXXX | | | | | | | | | |
| 05-CA-003 | Screening part | Yes | | 06/05/2013 | 9:45 | 178 | 85.9 | 27.3 | Yes | XXXXXXX | XXXXXXX | XXXXXXX |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_MR.

Note: NA = Not Available




Version: 021 Page: **78 of 96** 

# Listing 16.2.9.4: Vital Signs

| | | Evaluation | Have vital signs | Reason for | Vital signs | Vital signs | Height | Weight | Systolic BP | Diastolic BP | Pulse rate | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Visit | period | been evaluated? | non evaluation | evaluation date | evaluation time | (cm) | (kg) | (mmHg) | (mmHg) | (beats/min) | _ |
| PAT_PATNUMBE<br>R | VISIT_NAME | [Derived data] | VS_PRE_YN<br>VS_POST_YN | VS_PRE_YN_SP<br>VS_POST_YN_SP | VS_PRE_DATE<br>VS_POST_DATE | VS_PRE_TIME<br>VS_POST_TIME | | | VS_PRE_SBP<br>VS_POST_SBP | VS_PRE_DBP<br>VS_POST_SBP | VS_PRE_HR<br>VS_POST_HR | |
| 05-CA-001 | Screening<br>part 2 | Before injection | Yes | | 09/04/2011 | 12:00 | 175 | XX.X | 165 | 99 | 77 | |
| 05-CA-001 | Screening<br>part 2 | After injection | Yes | | 12/04/2011 | 10:00 | | | 129 | 93 | 60 | |
| 05-CA-002 | Visit 1 | Before injection | Yes | | 06/05/2013 | 9:45 | | XX.X | 147 | 68 | 76 | |
| 05-CA-002 | Visit 1 | After injection | No | XXXXXXXX | | | | | | | | |

Data Source Table: W\_PATIENT, W\_PATIENTVIS, W\_VS.

Note: NA = Not Available



Version: 021 Page: **79 of 96** 

# 11.2 Standard Tables




Version: 021 Page: **80 of 96** 

Table 14.1.1: Subject disposition

| POPULATION | STATISTIC | ALL<br>SUBJECT<br>S<br>(N=xx) |
|-----------------------------|-----------|-------------------------------|
| Screened subjects | n (%) | 99 (99.9) |
| Screen failures | n (%) | 99 (99.9) |
| Reason 1 | n (%) | 99 (99.9) |
| | n (%) | 99 (99.9) |
| Reason m | n (%) | 99 (99.9) |
| Enrolled subjects | n (%) | 99 (99.9) |
| Dosed subjects | n (%) | 99 (99.9) |
| Completed study subjects | n (%) | 99 (99.9) |
| Discontinued study subjects | n (%) | 99 (99.9) |
| Reason 1 | n (%) | 99 (99.9) |
| | n (%) | 99 (99.9) |
| Reason m | n (%) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: All percentages are based upon the number of screened subjects.




Version: 021 Page: **81 of 96** 

# **Table 14.1.4.1: Demographics – FAS Population**

| PARAMETER | | STATISTIC | FAS<br>(N=xx) |
|-------------|-----------|-----------|---------------|
| Age (years) | | n | 99 |
| | | Missing | 99 |
| | | Mean | 99.9 |
| | | S.D. | 99.9 |
| | | Median | 99.9 |
| | | Q1, Q3 | 99.9, 99.9 |
| | | Min, Max | 99, 99 |
| Ethnicity | Asian | n (%) | 99 (99.9) |
| | Black | n (%) | 99 (99.9) |
| | Caucasian | n (%) | 99 (99.9) |
| | Hispanic | n (%) | 99 (99.9) |
| | Other | n (%) | 99 (99.9) |
| | Missing | n (%) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: The denominator for the percentage is based on the number of subjects in the FAS population.




Version: 021 Page: **82 of 96** 

# Table 14.1.7.2/1: Study Drug Administration – Safety Population

| QUALITY CONTROL ON<br>THE FINAL PRODUCT | STATISTIC | SCREENING<br>PART 2<br>(N=xx) | VISIT 2<br>(N=xx) | VISIT 3<br>(N=xx) | VISIT 4<br>(N=xx) |
|---|---|---|---|---|---|
| Radiochemical purity (%) | n | 99 | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Notes: Acceptance criteria is radiochemical purity ≥ 90%.

N = total number of subjects in Safety population; n = number of subjects who received Annexin injection.




Version: 021 Page: **83 of 96** 

# Table 14.1.7.2/2: Study Drug Administration – Safety Population

| QUALITY CONTROL ON<br>THE FINAL PRODUCT | STATISTIC | SCREENING<br>PART 2<br>(N=xx) | VISIT 2<br>(N=xx) | VISIT 3<br>(N=xx) | VISIT 4<br>(N=xx) |
|---|---|---|---|---|---|
| Pre-injection total activity-dose in the syringe (MBq) | e n | 99 | 99 | 99 | 99 |
| 5)gc (24) | Missing | 99 | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 | 99, 99 |
| Post-injection residual activity-dose in the syringe (MBq) | e n | 99 | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: N = total number of subjects in Safety population; n = number of subjects who received Annexin injection.




Version: 021 Page: **84 of 96** 

# Table 14.1.7.2/3: Study Drug Administration – Safety Population

| QUALITY CONTROL ON<br>THE FINAL PRODUCT | STATISTIC | SCREENING<br>PART 2<br>(N=xx) | VISIT 2<br>(N=xx) | VISIT 3<br>(N=xx) | VISIT 4<br>(N=xx) |
|---|---|---|---|---|---|
| Actual dose in the syringe (MBq) | n | 99 | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 | 99, 99 |
| Volume of administered solution (mL) | n | 99 | 99 | 99 | 99 |
| | Missing | 99 | 99 | 99 | 99 |
| | Mean | 99.9 | 99.9 | 99.9 | 99.9 |
| | S.D. | 99.9 | 99.9 | 99.9 | 99.9 |
| | Median | 99.9 | 99.9 | 99.9 | 99.9 |
| | Q1, Q3 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 | 99.9, 99.9 |
| | Min, Max | 99, 99 | 99, 99 | 99, 99 | 99, 99 |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: N = total number of subjects in Safety population; n = number of subjects who received Annexin injection.




Version: 021 Page: **85 of 96** 

# Table 14.3.1.1: Overall Summary of Adverse Events – Safety Population

| ADVERSE EVENT CATEGORY | STATISTIC | SAFETY<br>(N=xx) |
|---|---|---|
| Treatment emergent AEs | n (%) [n. events] | 99 (99.9) [99] |
| Treatment emergent adverse drug reactions | n (%) [n. events] | 99 (99.9) [99] |
| Treatment emergent SAEs | n (%) [n. events] | 99 (99.9) [99] |
| Treatment emergent serious adverse drug reactions | n (%) [n. events] | 99 (99.9) [99] |
| Treatment emergent AEs leading to withdrawal | n (%) [n. events] | 99 (99.9) [99] |
| Treatment emergent AEs leading to death | n (%) [n. events] | 99 (99.9) [99] |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}

Note: Format is number of subjects (percent of subjects) [number of events].




Version: 021 Page: **86 of 96** 

# Table 14.3.1.2: Number (%) of Subjects Reporting Treatment Emergent Adverse Events by Primary System Organ Class and Preferred Term – Safety Population

| PRIMARY SYSTEM ORGAN CLASS<br>PREFERRED TERM | STATISTIC | SAFETY<br>(N=xx) |
|----------------------------------------------|-----------|------------------|
| Any adverse events | n (%) | 99 (99.9) |
| System organ class 1 | n (%) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) |
| | n (%) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) |
| System organ class | n (%) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) |
| | n (%) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) |
| System organ class m | n (%) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) |
| | n (%) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary

Name: MedDRA Version: 19.0

Notes: The denominator for the percentage is based on the number of subjects in the Safety population. Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT






Version: 021 Page: **87 of 96** 

# Table 14.3.1.3: Number (%) of Subjects Reporting Treatment Emergent Adverse Events by Severity – Safety Population

| PRIMARY SYSTEM<br>ORGAN CLASS<br>PREFERRED<br>TERM | Grade 1<br>(Mild) | Grade 2<br>(Modera<br>te) | Grade 3<br>(Severe) | Grade 4<br>(Threate<br>ning/dis<br>abling) | Grade 5<br>(Death) | Missing | Total |
|---|---|---|---|---|---|---|---|
| Any adverse events | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| ••• | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| ••• | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary

Name: MedDRA Version: 19.0

Notes: The denominator for the percentage is based on the number of subjects in the Safety population. Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT and the maximum CTC grade will be reported.






Version: 021 Page: **88 of 96** 

# Table 14.3.1.4: Number (%) of Subjects Reporting Treatment Emergent Adverse Drug Reactions by Severity – Safety Population

| PRIMARY SYSTEM ORGAN CLASS PREFERRED TERM | Grade 1<br>(Mild) | Grade 2<br>(Modera<br>te) | Grade 3<br>(Severe) | Grade 4<br>(Threate<br>ning/dis<br>abling) | Grade 5<br>(Death) | Missing | Total |
|---|---|---|---|---|---|---|---|
| Any adverse drug reactions | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| *** | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| *** | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| ••• | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary

Name: MedDRA Version: 19.0

Notes: The denominator for the percentage is based on the number of subjects in the Safety population. Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT and the maximum CTC grade will be reported.




Version: 021 Page: **89 of 96** 

Table 14.3.1.5: Number (%) of Subjects Reporting Treatment Emergent Serious Adverse Events by Primary System Organ Class and Preferred Term – Safety Population

| PRIMARY SYSTEM ORGAN CLASS<br>PREFERRED TERM | STATISTIC | SAFETY<br>(N=xx) |
|---|---|---|
| Any serious adverse events | n (%) | 99 (99.9) |
| System organ class 1 | n (%) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) |
| | n (%) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) |
| System organ class | n (%) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) |
| | n (%) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) |
| System organ class m | n (%) | 99 (99.9) |
| Preferred term 1 | n (%) | 99 (99.9) |
| | n (%) | 99 (99.9) |
| Preferred term m | n (%) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary

Name: MedDRA Version: 19.0

Notes: The denominator for the percentage is based on the number of subjects in the Safety population. Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT.






Version: 021 Page: **90 of 96** 

# Table 14.3.1.6: Number (%) of Subjects Reporting Treatment Emergent Serious Adverse Events by Severity – Safety Population

| PRIMARY SYSTEM ORGAN CLASS PREFERRED TERM | Grade 1<br>(Mild) | Grade 2<br>(Modera<br>te) | Grade 3<br>(Severe) | Grade 4<br>(Threate<br>ning/dis<br>abling) | Grade 5<br>(Death) | Missing | Total |
|---|---|---|---|---|---|---|---|
| Any serious adverse events | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| ••• | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| ••• | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary

Name: MedDRA Version: 19.0

Notes: The denominator for the percentage is based on the number of subjects in the Safety population. Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT and the maximum CTC grade will be reported.






Version: 021 Page: **91 of 96** 

# Table 14.3.1.7: Number (%) of Subjects Reporting Treatment Emergent Serious Adverse Drug Reactions by Severity – Safety Population

| PRIMARY SYSTEM ORGAN CLASS PREFERRED TERM | Grade 1<br>(Mild) | Grade 2<br>(Modera<br>te) | Grade 3<br>(Severe) | Grade 4<br>(Threate<br>ning/dis<br>abling) | Grade 5<br>(Death) | Missing | Total |
|---|---|---|---|---|---|---|---|
| Any serious adverse drug reactions | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| System organ class m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term 1 | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |
| Preferred term m | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) | 99 (99.9) |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary

Name: MedDRA Version: 19.0

Notes: The denominator for the percentage is based on the number of subjects in the Safety population. Subjects with more than one event within a particular SOC and PT will be counted only once for that SOC and PT and the maximum CTC grade will be reported.




Version: 021 Page: **92 of 96** 

# Table 14.3.2.1: Listing of Adverse Events with Outcome Death – Safety Population

| Subject ID | Age | Primary cause<br>of death | Date of study<br>drug<br>latest<br>injection | Time of study<br>drug<br>latest<br>injection | Date of<br>death | Time between study<br>drug<br>latest injection and<br>death (days) | Relationship<br>with study<br>treatment |
|---|---|---|---|---|---|---|---|
| 05-CA-001 | 82 | Heart Attack | 10/05/2012 | 11:30 | 17/05/2012 | 7 | Probable |
| 05-CA-002 | 88 | Aneurysm | 05/10/2012 | 12:38 | 08/10/2012 | 3 | Possible |
| 05-CA-003 | 71 | Tuberculosis | 15/07/2012 | 09:45 | 16/10/2012 | 1 | Unlikely |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets}




Version: 021 Page: **93 of 96** 

# Table 14.3.2.2: Listing of Serious Adverse Events – Safety Population

| Subject ID | Event description | Primary<br>system<br>organ<br>class | Preferred term | SAE<br>date | Study day<br>of onset<br>(days)# | Duration<br>(days) | SAE<br>criteria | Relationship<br>with study<br>treatment | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| 04-CA-001 | Vertigo | Ear and<br>labyrinth<br>disorders | Vertigo | 14/05/20<br>12 | 1 | <1 | 2, 3 | Unlikely | Resolved |
| 04-CA-002 | Fainting | Nervous<br>system<br>disorders | Syncope | 10/09/20<br>12 | 15 | <1 | 2 | Unlikely | Resolved<br>with<br>sequelae |
| 04-CA-003 | Internal<br>bleeding | Vascular<br>disorders | Internal<br>haemorrha<br>ge | 16/11/20<br>11 | 4 | 3 | 5 | Probable | Improved |
| | | ••• | | | | | | | |

Source: Data listings {Specify data listing number(s)} Analysis dataset: {Specify datasets} Dictionary name: MedDRA Version XX.X Note: SAE criteria: 1=Death, 2=Life-threatening, 3=Involved or prolonged hospitalization, 4=Congenital anomaly, 5=Persistent or significant disability or incapacity, 6=Significant from a medical standpoint.

<sup>\*</sup> Study day of onset is days since first annexin administration.


Version: 021 Page: **94 of 96** 

# 11.3 Standard Figures

The different lines on the figures should look different (e.g. dotted lines) rather than using different colours so that the lines can be distinguished when using a non-colour printer.




Version: 021 Page: **95 of 96** 

### 12 APPENDICES TO THE SAP TEMPLATE

### 12.1 Derived data

The following derived data will be calculated and included in the listings or in the tables:

### (1) Age

Subject age (years) will be derived as (first visit date - birth date)/365.25 and truncated to the largest integer that is less than or equal to the calculated result. Since birth date is truncated (i.e. only month and year will be filled in the eCRF), it will be approximated using "01" as value for the day.

### (2) **BMI**

BMI (kg/m²) will be automatically derived as [WEIGHT] (kg)/([HEIGHT](cm)/100)² and rounded to the nearest decimal.

### (3) Time from injection

Time from injection (min) will be derived as the difference between SPECT or SPECT/CT scan time and injection time [SP\_TIME/SPCT\_TIME - ANN\_TIME].

### (4) Adverse event duration

If the start and end dates of the adverse event are identical then "<1" day will be presented with the duration in hh:mm recorded in the eCRF if it is available. If times are available, the duration will be calculated as (end date/time - start date/time) and presented in days hh:mm. If at least one time is missing and if the duration is greater than 24 hours then it will be calculated as (end date - start date)+1 and presented in days. If the recorded end date is CONT. (for continuing), the end date will be listed as "ongoing" and the duration will be approximated as " $\geq$ (last attended visit date - start date)+1" day(s). If the start date or the end date are partial the duration will be presented as a superior inequality " $\geq$  xx" day(s) (i.e. " $\geq$ 2" where start date = 31JAN2004 and end date = FEB2004 or start date = JAN2004 and end date = 01FEB2004).

### (5) Study day of onset

If the start date of the adverse event is identical to the date of injection, then "1" day will be presented with the time to onset in hh:mm recorded in the eCRF if it is available. If the date of onset is greater than the date of injection then it will be calculated as (start date - injection date+1) and presented in days. If the date of onset precedes the date of injection the study day will be calculated as (start date - injection date). If the start date is partial, the time since injection will be presented as a superior inequality (i.e. for an AE started in FEB2004 after the injection performed on 31JAN2004, the delay of onset will be "≥2" days).




Version: 021 Page: **96 of 96** 

# 12.2 SAS programs

This section provides the SAS programs related to the statistical tests specified in the statistical methods section 6. All computer output from SAS statistical programs used as a basis for extracted results should be retained for review by Responsible of statistical analysis.



**Proc Format** 

**Proc Print** 

**Proc Sort** 

Proc SQL

**Proc Transpose** 

### 2 Descriptive statistics

Proc Corr

Proc Freq

**Proc Means** 

Proc Tabulate

### 3 Test statistics

Proc GLM

Proc Mixed

Proc Ttest

**Proc Univariate** 

### 4 Graphs

**Proc Boxplot** 

**Proc Sgplot**